CLINICAL TRIAL: NCT04263142
Title: A Two-Part, Randomized, Open-Label, Single Dose, Crossover Clinical Trial to Assess the Relative Bioavailability of a Tablet Compared to a Capsule of GSK3640254 and to Assess the Effect of Food on the GSK3640254 Tablet in Healthy Participants
Brief Title: A Relative Bioavailability and Food-Effect Study of GSK3640254 Tablet and Capsule Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 213567
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: HIV Infections
Keywords: Healthy participants; GSK3640254; Human immunodeficiency virus; Relative Bioavailability
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — GSK3640254

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned to 1 of 2 treatment sequences (AB or BA) in Part 1 and 1 of 3 treatment sequences (CDE, DEC, or ECD) in Part 2.
Masking Description: This is an open label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Treatment AB (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment A- Reference), capsules, orally under moderate fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment B- Test), tablets, orally under moderate fat conditions on Day 1 in second intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet; Drug: GSK3640254 Capsule
- Part 1: Treatment BA (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment B- Test), tablets, orally under moderate fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment A- Reference), capsules, orally under moderate fat conditions on Day 1 in second intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet; Drug: GSK3640254 Capsule
- Part 2: Treatment CDE (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment C- Test), tablets, orally under moderate fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment D- Reference), tablets, orally under fasted conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment E- Test), tablets, orally under high fat conditions on Day 1 in third intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet
- Part 2: Treatment DEC (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment D- Reference), tablets, orally under fasted conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment E- Test), tablets, orally under high fat conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment C- Test), tablets, orally under moderate fat conditions on Day 1 in third intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet
- Part 2: Treatment ECD (Experimental): Participants will receive a single dose of GSK3640254 200 mg (Treatment E- Test), tablets, orally under high fat conditions on Day 1 in first intervention period; followed by GSK3640254 200 mg (Treatment C- Test), tablets, orally under moderate fat conditions on Day 1 in second intervention period; followed by GSK3640254 200 mg (Treatment D- Reference), tablets, orally under fasted conditions on Day 1 in third intervention period. There will be at least 7 days wash out period between each dose of study intervention.
  Interventions: Drug: GSK3640254 Tablet

INTERVENTIONS:
Drug: GSK3640254 Tablet — GSK3640254 tablets will contain mesylate salt with a unit dose of 100 mg (2x100 mg) and will be administered orally.
Drug: GSK3640254 Capsule — GSK3640254 capsules will contain mesylate salt with a unit dose of 100 mg (2x100 mg) and will be administered orally.
  Arms: Part 1: Treatment AB; Part 1: Treatment BA

SUMMARY:
This is an open-label, 2 part, single-dose and crossover study conducted to assess the relative bioavailability of a tablet compared to a capsule of GSK3640254 and to assess the effect of food on the GSK3640254 tablet in healthy participants. This study will also evaluate the effect of food (fasted, moderate fat meal, and high fat meal) on the pharmacokinetics of the GSK3640254 mesylate tablet formulation. In Part 1, participants will be randomly assigned to 1 of 2 treatment sequences (AB or BA) in two sequential treatment periods; and in Part 2, participants will be randomly assigned to 1 of 3 treatment sequences (CDE, DEC, or ECD) in three sequential treatment periods. Participants will be randomized to receive a single dose of GSK3640254 200 milligram (mg) capsules under moderate fat conditions and GSK3640254 200 mg tablets under moderate fat, fasted and high fat conditions in each treatment period. Approximately 30 participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria

* Participants must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and ECG).
* Body weight >=50.0 kilogram (kg) (110 pounds [lbs]) for men and >=45.0 kg (99 lbs) for women and body mass index within the range 18.5 to 31.0 kg per square meter (kg/m^2) (inclusive).
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants: Males shall not engage in intercourse while confined in the clinic. There is no need for an extended period of double barrier use or prolonged abstinence after study discharge. Female participants: 1. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least 1 of the following conditions applies: a. not a woman of childbearing potential (WOCBP); or Is a WOCBP and using a nonhormonal contraceptive method that is highly effective, with a failure rate of <1 percent (%), for 28 days before intervention, during the intervention period, and for at least 28 days after the last dose of study intervention. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention. 2. A WOCBP must have a negative highly sensitive serum pregnancy test at Screening and Day -1. 3. Additional requirements for pregnancy testing during and after study intervention.
* The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions.

Exclusion Criteria

* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A pre-existing condition interfering with normal gastrointestinal (GI) anatomy or motility (example [e.g.], gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study intervention or render the participant unable to take oral study intervention.
* Prior cholecystectomy surgery (prior appendectomy is acceptable).
* Any history of significant underlying psychiatric disorder, including, but not limited to, schizophrenia, bipolar disorder with or without psychotic symptoms, other psychotic disorders, or schizotypal (personality) disorder.
* Any history of major depressive disorder with or without suicidal features, or anxiety disorders that required medical intervention (pharmacologic or not) such as hospitalization or other inpatient treatment and/or chronic (>6 months) outpatient treatment. Participants with other conditions such as adjustment disorder or dysthymia that have required shorter term medical therapy (<6 months) without inpatient treatment and are currently well-controlled clinically or resolved may be considered for entry after discussion and agreement with the Medical Monitor.
* Any pre-existing physical or other psychiatric condition (including alcohol or drug abuse), which, in the opinion of the investigator (with or without psychiatric evaluation), could interfere with the participant's ability to comply with the dosing schedule and protocol evaluations or which might compromise the safety of the participant.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* Presence of hepatitis B surface antigen at Screening or within 3 months prior to starting study intervention.
* Positive hepatitis C antibody test result at Screening or within 3 months prior to starting study intervention and positive on reflex to hepatitis C ribonucleic acid (RNA).
* Positive Human immunodeficiency virus (HIV)-1 and -2 antigen/antibody immunoassay at Screening.
* ALT >1.5 times upper limit of normal (ULN). A single repeat of ALT is allowed within a single Screening period to determine eligibility.
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* Any acute laboratory abnormality at Screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at Screening, with the exception of creatine phosphokinase (CPK) and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT (described above), will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor. A single repeat of any laboratory abnormality is allowed within a single Screening period to determine eligibility.
* A positive test result for drugs of abuse (including marijuana), alcohol, or cotinine (indicating active current smoking) at Screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or nonprescription drugs including vitamins, herbal and dietary supplements (including Saint John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study intervention and for the duration of the study.
* Treatment with any vaccine within 30 days prior to receiving study intervention.
* Unwillingness to abstain from excessive consumption of any food or drink containing grapefruit and grapefruit juice, Seville oranges, blood oranges, or pomelos or their fruit juices within 7 days prior to the first dose of study intervention(s) until the end of the study.
* Participation in another concurrent clinical study or prior clinical study (with the exception of imaging trials) prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the study intervention (whichever is longer).
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Any positive (abnormal) response confirmed by the investigator on a screening clinician- or qualified designee-administered Columbia Suicide Severity Rating Scale (C-SSRS).
* Any significant arrhythmia or ECG finding (e.g., prior myocardial infarction in the past 3 months, symptomatic bradycardia, non-sustained or sustained atrial arrhythmias, non-sustained or sustained ventricular tachycardia, second-degree atrioventricular block Mobitz Type II, third-degree atrioventricular block, complete heart block, or conduction abnormality) which, in the opinion of the investigator or Medical Monitor, will interfere with the safety for the individual participant.
* Exclusion criteria for Screening ECG (a single repeat is allowed for eligibility determination): Heart rate: <50 or >100 beats per minute and QTcF interval: >450 millisecond.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 units. One unit is equivalent to 8 grams of alcohol: a half pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine, or 1 (25 mL) measure of spirits.
* Unable to refrain from tobacco or nicotine-containing products within 3 months prior to Screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Johnson M, Pene Dumitrescu T, Joshi SR, Mathew A, Bainbridge V, Zhan J, Lataillade M. Relative Bioavailability and Food Effect of GSK3640254 Tablet and Capsule Formulations in Healthy Participants. Clin Pharmacol Drug Dev. 2022 May;11(5):632-639. doi: 10.1002/cpdd.1051. Epub 2022 Jan 7. PMID 34995417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-part, randomized, single dose cross-over study conducted at a single center in the United States to assess the relative bioavailability and food effect of GSK3640254 tablet and capsule formulations in healthy participants.
Pre-assignment Details: A total of 39 participants were enrolled in Part 1 (18 participants) and Part 2 (21 participants) of the study.
Groups:
- Part 1: Treatment Sequence AB: Participants were administered a single dose of GSK3640254 200 milligram (mg) capsules (Treatment A-reference), orally under moderate fat conditions on Day 1 in Period 1, followed by GSK3640254 200 mg tablets (Treatment B- test), orally under moderate fat conditions on Day 1 in Period 2. There was a wash out period of at least 7 days between each dose of study intervention.
- Part 1: Treatment Sequence BA: Participants were administered a single dose of GSK3640254 200 mg tablets (Treatment B-test), orally under moderate fat conditions on Day 1 in Period 1, followed by GSK3640254 200 mg capsules (Treatment A-reference), orally under moderate fat conditions on Day 1 in Period 2. There was a wash out period of at least 7 days between each dose of study intervention.
- Part 2: Treatment Sequence CDE: Participants were administered a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment C-test) on Day 1 in Period 1, followed by GSK3640254 200 mg tablets, orally under fasted conditions (Treatment D-reference) on Day 1 in Period 2, followed by GSK3640254 200 mg tablets, orally under high fat conditions (Treatment E-test) on Day 1 in Period 3. There was a wash out period of at least 7 days between each dose of study intervention.
- Part 2: Treatment Sequence DEC: Participants were administered a single dose of GSK3640254 200 mg tablets, orally under fasted conditions (Treatment D-reference) on Day 1 in Period 1, followed by GSK3640254 200 mg tablets, orally under high fat conditions (Treatment E-test) on Day 1 in Period 2, followed by GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment C-test) on Day 1 in Period 3. There was a wash out period of at least 7 days between each dose of study intervention.
- Part 2: Treatment Sequence ECD: Participants were administered a single dose of GSK3640254 200 mg tablets, orally under high fat conditions (Treatment E-test) on Day 1 in Period 1; followed by GSK3640254 200 mg tablets, orally under moderate fat conditions (Treatment C-test) on Day 1 in Period 2; followed by GSK3640254 200 mg tablets, orally under fasted conditions (Treatment D-reference) on Day 1 in Period 3. There was a wash out period of at least 7 days between each dose of study intervention.
Period: Part 1 Period 1 (Day 1)
Arm/Group | Part 1: Treatment Sequence AB | Part 1: Treatment Sequence BA | Part 2: Treatment Sequence CDE | Part 2: Treatment Sequence DEC | Part 2: Treatment Sequence ECD
Started | 9 | 9 | 0 | 0 | 0
Completed | 9 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 1 Period 2 (Up to Day 5)
Arm/Group | Part 1: Treatment Sequence AB | Part 1: Treatment Sequence BA | Part 2: Treatment Sequence CDE | Part 2: Treatment Sequence DEC | Part 2: Treatment Sequence ECD
Started | 9 | 9 | 0 | 0 | 0
Completed | 9 | 9 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2 Period 1 (Day 1)
Arm/Group | Part 1: Treatment Sequence AB | Part 1: Treatment Sequence BA | Part 2: Treatment Sequence CDE | Part 2: Treatment Sequence DEC | Part 2: Treatment Sequence ECD
Started | 0 | 0 | 7 | 7 | 7
Completed | 0 | 0 | 7 | 7 | 6
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Part 2 Period 2 (Day 1)
Arm/Group | Part 1: Treatment Sequence AB | Part 1: Treatment Sequence BA | Part 2: Treatment Sequence CDE | Part 2: Treatment Sequence DEC | Part 2: Treatment Sequence ECD
Started | 0 | 0 | 7 | 7 | 6
Completed | 0 | 0 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Period: Part 2 Period 3 (Up to Day 5)
Arm/Group | Part 1: Treatment Sequence AB | Part 1: Treatment Sequence BA | Part 2: Treatment Sequence CDE | Part 2: Treatment Sequence DEC | Part 2: Treatment Sequence ECD
Started | 0 | 0 | 7 | 7 | 5
Completed | 0 | 0 | 7 | 7 | 5
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Treatment Sequence AB | Part 1: Treatment Sequence BA | Part 2: Treatment Sequence CDE | Part 2: Treatment Sequence DEC | Part 2: Treatment Sequence ECD | Total
Number analyzed (Participants) | 9 | 9 | 7 | 7 | 7 | 39
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  19 to 64 years | 9 | 9 | 7 | 7 | 7 | 39
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 5 | 14
  Male | 7 | 6 | 4 | 6 | 2 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 2 | 3 | 2 | 4 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  White-Arabic/North African Heritage | 0 | 1 | 0 | 0 | 0 | 1
  White-White/Caucasian/European Heritage | 4 | 5 | 4 | 5 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0 to Inf]) for GSK3640254-Part 1
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population comprised of all participants who underwent plasma PK sampling and had evaluable PK parameters estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Groups:
- Part 1: GSK3640254 200 mg Capsules: Participants were administered a single dose of GSK3640254 200 mg capsules, orally under moderate fat conditions on Day 1 in Period 1 or 2.
- Part 1: GSK3640254 200 mg Tablets: Participants were administered a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions on Day 1 in Period 1 or 2.
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Hours*microgram per milliliter | 36.94 (42.7) | 36.88 (40.3)
Statistical Analysis 1: Comparison: Part 1: GSK3640254 200 mg Capsules vs Part 1: GSK3640254 200 mg Tablets; Test type: Other; Ratio = 0.998, 90% CI 2-sided [0.9263 to 1.0757] — Analysis was performed using analysis of variance (ANOVA) with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter AUC(0-inf). Ratio of GSK3640254 200 mg tablets/capsules

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Time t (AUC[0 to t]) for GSK3640254-Part 1
Description: Blood samples were collected at indicated time points for PK analysis. PK parameters were calculated using standard non-compartmental analysis.
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Hours*microgram per milliliter | 33.72 (41.1) | 33.80 (40.2)
Statistical Analysis 1: Comparison: Part 1: GSK3640254 200 mg Capsules vs Part 1: GSK3640254 200 mg Tablets; Test type: Other; Ratio = 1.002, 90% CI 2-sided [0.9321 to 1.0781] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter AUC(0-t). Ratio of GSK3640254 200 mg tablets/capsules

3. Primary Outcome: Maximum Observed Concentration (Cmax) for GSK3640254-Part 1
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Microgram per milliliter | 1.201 (33.4) | 1.313 (45.3)
Statistical Analysis 1: Comparison: Part 1: GSK3640254 200 mg Capsules vs Part 1: GSK3640254 200 mg Tablets; Test type: Other; Ratio = 1.093, 90% CI 2-sided [0.9885 to 1.2080] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter Cmax. Ratio of GSK3640254 200 mg tablets/capsules

4. Primary Outcome: Time of Maximum Observed Concentration for GSK3640254-Part 1
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Hours | 5.000 [3.00 to 12.00] | 4.000 [2.50 to 6.00]

5. Primary Outcome: AUC(0 to Inf) for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Groups:
- Part 2: GSK3640254 200 mg Tablet (Moderate Fat): Participants were administered a single dose of GSK3640254 200 mg tablets, orally under moderate fat conditions on Day 1 in Period 1, 2 or 3.
- Part 2: GSK3640254 200 mg Tablet (Fasted): Participants were administered a single dose of GSK3640254 200 mg tablets, orally under fasted conditions on Day 1 in Period 1, 2 or 3.
- Part 2: GSK3640254 200 mg Tablet (High Fat): Participants were administered a single dose of GSK3640254 200 mg tablets, orally under high fat conditions on Day 1 in Period 1, 2 or 3.
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 10 | 21
Hours*micrograms per milliliter | 41.00 (42.2) | 13.46 (58.2) | 36.92 (35.9)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 200 mg Tablet (Moderate Fat) vs Part 2: GSK3640254 200 mg Tablet (Fasted); Test type: Other; Ratio = 2.926, 90% CI 2-sided [2.3703 to 3.6107] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter AUC(0-inf). Ratio of GSK3640254 200 mg tablet (moderate fat)/(fasted)
Statistical Analysis 2: Comparison: Part 2: GSK3640254 200 mg Tablet (Fasted) vs Part 2: GSK3640254 200 mg Tablet (High Fat); Test type: Other; Ratio = 2.594, 90% CI 2-sided [2.1003 to 3.2038] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter AUC(0-inf). Ratio of GSK3640254 200 mg tablet (high fat)/(fasted)

6. Primary Outcome: AUC(0 to t) for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*micrograms per milliliter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 13 | 21
Hours*micrograms per milliliter | 37.91 (41.5) | 11.37 (65.6) | 34.08 (34.9)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 200 mg Tablet (Moderate Fat) vs Part 2: GSK3640254 200 mg Tablet (Fasted); Test type: Other; Ratio = 3.146, 90% CI 2-sided [2.5925 to 3.8178] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter AUC(0-t). Ratio of GSK3640254 200 mg tablet (moderate fat)/(fasted)
Statistical Analysis 2: Comparison: Part 2: GSK3640254 200 mg Tablet (Fasted) vs Part 2: GSK3640254 200 mg Tablet (High Fat); Test type: Other; Ratio = 2.785, 90% CI 2-sided [2.2943 to 3.3807] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter AUC(0-t). Ratio of GSK3640254 200 mg tablet (high fat)/(fasted)

7. Primary Outcome: Cmax for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 13 | 21
Micrograms per milliliter | 1.425 (35.6) | 0.3544 (84.4) | 1.082 (38.6)
Statistical Analysis 1: Comparison: Part 2: GSK3640254 200 mg Tablet (Moderate Fat) vs Part 2: GSK3640254 200 mg Tablet (Fasted); Test type: Other; Ratio = 4.101, 90% CI 2-sided [3.2442 to 5.1830] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter Cmax. Ratio of GSK3640254 200 mg tablet (moderate fat)/(fasted)
Statistical Analysis 2: Comparison: Part 2: GSK3640254 200 mg Tablet (Fasted) vs Part 2: GSK3640254 200 mg Tablet (High Fat); Test type: Other; Ratio = 3.080, 90% CI 2-sided [2.4359 to 3.8935] — Analysis was performed using ANOVA with treatment, period, and sequence as fixed effects and participant as a random effect on the natural log-transformed parameter Cmax. Ratio of GSK3640254 200 mg tablet (high fat)/(fasted)

8. Primary Outcome: Time of Maximum Observed Concentration for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 13 | 21
Hours | 5.000 [2.00 to 8.00] | 4.000 [2.03 to 24.00] | 5.000 [1.50 to 12.00]

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)-Part 1
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment.
Time Frame: Up to Day 12
Population: Safety Population comprised of all participants who received at least 1 dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Participants
  AEs | 0 | 1
  SAEs | 0 | 0

10. Secondary Outcome: Number of Participants With AEs and SAEs-Part 2
Description: as for outcome 9
Time Frame: Up to Day 19
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Participants
  AEs | 0 | 0 | 5
  SAEs | 0 | 0 | 0

11. Secondary Outcome: Absolute Values of Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets-Part 1
Description: Blood samples were collected for the assessment of following hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelets.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles)
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
10^9 cells per liter
  Basophils; Baseline; n=18, 18 | 0.032 (0.0134) | 0.032 (0.0134)
  Basophils; Day 2; n=18, 18 | 0.030 (0.0137) | 0.030 (0.077)
  Basophils; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Basophils; Day 5; n=9, 9 | 0.027 (0.0071) | 0.030 (0.0166)
  Eosinophils; Baseline; n=18, 18 | 0.100 (0.0832) | 0.100 (0.0832)
  Eosinophils; Day 2; n=18, 18 | 0.116 (0.0911) | 0.122 (0.1101)
  Eosinophils; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Eosinophils; Day 5; n=9, 9 | 0.133 (0.1227) | 0.118 (0.0769)
  Lymphocytes; Baseline; n=18, 18 | 1.617 (0.3975) | 1.617 (0.3975)
  Lymphocytes; Day 2; n=18, 18 | 1.726 (0.3852) | 1.744 (0.4791)
  Lymphocytes; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Lymphocytes; Day 5; n=9, 9 | 1.639 (0.3536) | 2.074 (0.6328)
  Monocytes; Baseline; n=18, 18 | 0.403 (0.0859) | 0.403 (0.0859)
  Monocytes; Day 2; n=18, 18 | 0.409 (0.0955) | 0.412 (0.1379)
  Monocytes; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Monocytes; Day 5; n=9, 9 | 0.386 (0.1100) | 0.411 (0.1071)
  Neutrophils; Baseline; n=18, 18 | 3.406 (1.0436) | 3.406 (1.0436)
  Neutrophils; Day 2; n=18, 18 | 2.925 (0.6617) | 2.723 (0.9257)
  Neutrophils; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Neutrophils; Day 5; n=9, 9 | 2.864 (0.7372) | 3.108 (0.5724)
  Platelets; Baseline; n=18, 18 | 232.5 (43.58) | 232.5 (43.58)
  Platelets; Day 2; n=18, 18 | 238.2 (49.37) | 241.5 (48.56)
  Platelets; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Platelets; Day 5; n=9, 9 | 267.1 (52.86) | 231.4 (38.51)

12. Secondary Outcome: Absolute Values for Erythrocytes Count-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocytes count.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
10^12 cells per liter
  Baseline; n=18, 18 | 4.801 (0.4605) | 4.801 (0.4605)
  Day 2; n=18, 18 | 4.937 (0.4896) | 4.983 (0.5010)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 5.009 (0.4786) | 5.061 (0.3888)

13. Secondary Outcome: Absolute Values for Hemoglobin-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: hemoglobin.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Grams per liter
  Baseline; n=18, 18 | 142.2 (13.46) | 142.2 (13.46)
  Day 2; n=18, 18 | 146.4 (13.74) | 148.3 (14.29)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 150.3 (15.74) | 150.3 (13.13)

14. Secondary Outcome: Absolute Values for Hematocrit-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: hematocrit.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Proportion of red blood cells in blood
  Baseline; n=18, 18 | 0.4252 (0.03485) | 0.4252 (0.03485)
  Day 2; n=18, 18 | 0.4346 (0.03935) | 0.4405 (0.03885)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 0.4410 (0.04004) | 0.4430 (0.03266)

15. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Volume-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocyte mean corpuscular volume.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Femtoliters
  Baseline; n=18, 18 | 88.80 (4.887) | 88.80 (4.887)
  Day 2; n=18, 18 | 88.21 (4.480) | 88.61 (4.363)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 88.17 (4.532) | 87.63 (4.971)

16. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Hemoglobin-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocyte mean corpuscular hemoglobin.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Picograms
  Baseline; n=18, 18 | 29.68 (1.858) | 29.68 (1.858)
  Day 2; n=18, 18 | 29.69 (1.740) | 29.83 (1.772)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 30.08 (1.737) | 29.74 (1.938)

17. Secondary Outcome: Absolute Values of Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets-Part 2
Description: as for outcome 11
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
10^9 cells per liter
  Basophils; Baseline; n=20, 19, 21 | 0.042 (0.0260) | 0.042 (0.0260) | 0.042 (0.0260)
  Basophils; Day 2; n=20, 19, 21 | 0.041 (0.0276) | 0.040 (0.0200) | 0.043 (0.0215)
  Basophils; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Basophils; Day 5; n=7, 5, 7 | 0.047 (0.0287) | 0.036 (0.0167) | 0.049 (0.0219)
  Eosinophils; Baseline; n=20, 19, 21 | 0.141 (0.0879) | 0.141 (0.0879) | 0.141 (0.0879)
  Eosinophils; Day 2; n=20, 19, 21 | 0.136 (0.0922) | 0.135 (0.0837) | 0.150 (0.1109)
  Eosinophils; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Eosinophils; Day 5; n=7, 5, 7 | 0.146 (0.1050) | 0.090 (0.0374) | 0.151 (0.0915)
  Lymphocytes; Baseline; n=20, 19, 21 | 1.650 (0.4926) | 1.650 (0.4926) | 1.650 (0.4926)
  Lymphocytes; Day 2; n=20, 19, 21 | 1.576 (0.3410) | 1.684 (0.4939) | 1.583 (0.3748)
  Lymphocytes; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Lymphocytes; Day 5; n=7, 5, 7 | 1.806 (0.3577) | 1.472 (0.2765) | 1.923 (0.4442)
  Monocytes; Baseline; n=20, 19, 21 | 0.469 (0.1445) | 0.469 (0.1445) | 0.469 (0.1445)
  Monocytes; Day 2; n=20, 19, 21 | 0.446 (0.1589) | 0.449 (0.1171) | 0.446 (0.1553)
  Monocytes; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Monocytes; Day 5; n=7, 5, 7 | 0.530 (0.1788) | 0.422 (0.0669) | 0.504 (0.1130)
  Neutrophils; Baseline; n=20, 19, 21 | 3.246 (1.0719) | 3.246 (1.0719) | 3.246 (1.0719)
  Neutrophils; Day 2; n=20, 19, 21 | 2.908 (1.1660) | 2.904 (0.8595) | 2.947 (1.0824)
  Neutrophils; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Neutrophils; Day 5; n=7, 5, 7 | 2.464 (0.9204) | 3.472 (0.8987) | 3.877 (1.4452)
  Platelets; Baseline; n=20, 19, 21 | 259.9 (63.91) | 259.9 (63.91) | 259.9 (63.91)
  Platelets; Day 2; n=20, 19, 21 | 284.2 (55.70) | 270.6 (60.80) | 281.3 (59.88)
  Platelets; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Platelets; Day 5; n=7, 5, 7 | 255.9 (47.27) | 272.4 (77.61) | 291.3 (48.52)

18. Secondary Outcome: Absolute Values for Erythrocytes Count-Part 2
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocytes count.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
10^12 cells per liter
  Baseline; n=20, 19, 21 | 4.613 (0.5680) | 4.613 (0.5680) | 4.613 (0.5680)
  Day 2; n=20, 19, 21 | 4.893 (0.5814) | 4.899 (0.5878) | 4.850 (0.5900)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 4.941 (0.6086) | 4.424 (0.6683) | 4.957 (0.6309)

19. Secondary Outcome: Absolute Values for Hemoglobin-Part 2
Description: Blood samples were collected for the assessment of following hematology parameter: hemoglobin.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Grams per liter
  Baseline; n=20, 19, 21 | 134.0 (15.37) | 134.0 (15.37) | 134.0 (15.37)
  Day 2; n=20, 19, 21 | 140.6 (15.83) | 141.1 (16.19) | 140.0 (15.37)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 146.9 (14.14) | 124.2 (15.74) | 142.7 (14.42)

20. Secondary Outcome: Absolute Values for Hematocrit-Part 2
Description: Blood samples were collected for the assessment of following hematology parameter: hematocrit.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Proportion of red blood cells in blood
  Baseline; n=20, 19, 21 | 0.4010 (0.03876) | 0.4010 (0.03876) | 0.4010 (0.03876)
  Day 2; n=20, 19, 21 | 0.4207 (0.03989) | 0.4219 (0.04146) | 0.4176 (0.03777)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 0.4337 (0.03499) | 0.3786 (0.04858) | 0.4216 (0.03917)

21. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Volume-Part 2
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocyte mean corpuscular volume.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Femtoliters
  Baseline; n=20, 19, 21 | 86.98 (5.931) | 86.98 (5.931) | 86.98 (5.931)
  Day 2; n=20, 19, 21 | 86.37 (5.934) | 86.52 (6.038) | 86.57 (5.867)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 88.47 (8.285) | 85.86 (4.453) | 85.41 (4.401)

22. Secondary Outcome: Absolute Values for Erythrocyte Mean Corpuscular Hemoglobin-Part 2
Description: as for outcome 16
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Picograms
  Baseline; n=20, 19, 21 | 29.05 (2.499) | 29.05 (2.499) | 29.05 (2.499)
  Day 2; n=20, 19, 21 | 28.87 (2.415) | 28.92 (2.449) | 28.99 (2.411)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 29.96 (3.365) | 28.14 (1.394) | 28.93 (1.962)

23. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets-Part 1
Description: Blood samples were collected for the assessment of following hematology parameters: basophils, eosinophils, lymphocytes, monocytes, neutrophils and platelets. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
10^9 cells per liter
  Basophils; Day 2; n=18, 18 | -0.002 (0.0092) | -0.002 (0.0092)
  Basophils; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Basophils; Day 5; n=9, 9 | -0.002 (0.0083) | -0.004 (0.0073)
  Eosinophils; Day 2; n=18, 18 | 0.016 (0.0322) | 0.022 (0.0387)
  Eosinophils; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Eosinophils; Day 5; n=9, 9 | 0.022 (0.0441) | 0.029 (0.0462)
  Lymphocytes; Day 2; n=18, 18 | 0.109 (0.2237) | 0.127 (0.2350)
  Lymphocytes; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Lymphocytes; Day 5; n=9, 9 | 0.082 (0.2124) | 0.398 (0.3721)
  Monocytes; Day 2; n=18, 18 | 0.006 (0.0581) | 0.008 (0.1164)
  Monocytes; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Monocytes; Day 5; n=9, 9 | -0.009 (0.0821) | -0.001 (0.0637)
  Neutrophils; Day 2; n=18, 18 | -0.481 (0.7029) | -0.683 (0.8597)
  Neutrophils; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Neutrophils; Day 5; n=9, 9 | -0.291 (0.5628) | 0.549 (0.7398)
  Platelets; Day 2; n=18, 18 | 5.7 (21.18) | 9.0 (18.89)
  Platelets; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Platelets; Day 5; n=9, 9 | 20.8 (15.16) | 12.8 (22.55)

24. Secondary Outcome: Change From Baseline in Erythrocytes Count-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocytes count. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
10^12 cells per liter
  Day 2; n=18, 18 | 0.136 (0.2431) | 0.182 (0.2052)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 0.253 (0.2320) | 0.214 (0.1729)

25. Secondary Outcome: Change From Baseline in Hemoglobin-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: hemoglobin. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Grams per liter
  Day 2; n=18, 18 | 4.2 (7.11) | 6.1 (6.69)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 8.7 (7.66) | 7.6 (6.04)

26. Secondary Outcome: Change From Baseline in Hematocrit-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: hematocrit. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Proportion of red blood cells in blood
  Day 2; n=18, 18 | 0.0094 (0.02265) | 0.0153 (0.01912)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 0.0189 (0.02196) | 0.0147 (0.01362)

27. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocyte mean corpuscular volume. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Femtoliters
  Day 2; n=18, 18 | -0.59 (0.984) | -0.19 (1.050)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | -0.84 (0.911) | -0.96 (0.592)

28. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin-Part 1
Description: Blood samples were collected for the assessment of following hematology parameter: erythrocyte mean corpuscular hemoglobin. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Picograms
  Day 2; n=18, 18 | 0.01 (0.344) | 0.14 (0.365)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 0.26 (0.343) | 0.20 (0.439)

29. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelets-Part 2
Description: as for outcome 23
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
10^9 cells per liter
  Basophils; Day 2; n=20, 19, 21 | -0.001 (0.0107) | -0.003 (0.0129) | 0.001 (0.0128)
  Basophils; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Basophils; Day 5; n=7, 5, 7 | 0.000 (0.0100) | 0.006 (0.0114) | 0.000 (0.0129)
  Eosinophils; Day 2; n=20, 19, 21 | 0.001 (0.0424) | -0.006 (0.0519) | 0.009 (0.0464)
  Eosinophils; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Eosinophils; Day 5; n=7, 5, 7 | 0.007 (0.0423) | -0.030 (0.0738) | -0.009 (0.0402)
  Lymphocytes; Day 2; n=20, 19, 21 | -0.073 (0.2828) | 0.006 (0.3097) | -0.068 (0.2313)
  Lymphocytes; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Lymphocytes; Day 5; n=7, 5, 7 | 0.257 (0.2146) | -0.010 (0.1454) | -0.024 (0.4172)
  Monocytes; Day 2; n=20, 19, 21 | -0.028 (0.1055) | -0.022 (0.0978) | -0.022 (0.1272)
  Monocytes; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Monocytes; Day 5; n=7, 5, 7 | 0.024 (0.1081) | 0.000 (0.1058) | 0.034 (0.1509)
  Neutrophils; Day 2; n=20, 19, 21 | -0.326 (0.7627) | -0.336 (0.7377) | -0.300 (0.7173)
  Neutrophils; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Neutrophils; Day 5; n=7, 5, 7 | -0.216 (0.6986) | 0.154 (0.8131) | 0.134 (1.1111)
  Platelets; Day 2; n=20, 19, 21 | 21.6 (30.53) | 9.4 (25.64) | 21.4 (26.82)
  Platelets; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Platelets; Day 5; n=7, 5, 7 | 38.0 (26.03) | -5.8 (28.08) | -1.1 (30.28)

30. Secondary Outcome: Change From Baseline in Erythrocytes Count-Part 2
Description: as for outcome 24
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
10^12 cells per liter
  Day 2; n=20, 19, 21 | 0.256 (0.1751) | 0.247 (0.2564) | 0.237 (0.1682)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 0.231 (0.1520) | 0.172 (0.1678) | 0.077 (0.2276)

31. Secondary Outcome: Change From Baseline in Hemoglobin-Part 2
Description: as for outcome 25
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Grams per liter
  Day 2; n=20, 19, 21 | 6.5 (4.96) | 6.3 (7.39) | 6.0 (4.21)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 7.0 (3.11) | 4.2 (5.50) | 2.4 (5.32)

32. Secondary Outcome: Change From Baseline in Hematocrit-Part 2
Description: as for outcome 26
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Proportion of red blood cells in blood
  Day 2; n=20, 19, 21 | 0.0187 (0.01477) | 0.0182 (0.02179) | 0.0166 (0.01313)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 0.0179 (0.01378) | 0.0106 (0.01731) | 0.0046 (0.01855)

33. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume-Part 2
Description: as for outcome 27
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Femtoliters
  Day 2; n=20, 19, 21 | -0.35 (0.841) | -0.28 (0.897) | -0.41 (0.774)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | -0.06 (1.124) | -0.02 (1.103) | -0.33 (0.834)

34. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Hemoglobin-Part 2
Description: as for outcome 28
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Picograms
  Day 2; n=20, 19, 21 | -0.05 (0.330) | -0.05 (0.276) | -0.06 (0.356)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 0.10 (0.365) | 0.18 (0.536) | 0.13 (0.553)

35. Secondary Outcome: Absolute Values for Chemistry Parameters: Creatinine, Total Bilirubin, Direct Bilirubin and Urate-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: creatinine, total bilirubin, direct bilirubin and urate.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Micromoles per liter
  Creatinine; Baseline; n=18, 18 | 78.68 (15.983) | 78.68 (15.983)
  Creatinine; Day 2; n=18, 18 | 80.87 (15.104) | 80.11 (14.243)
  Creatinine; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Creatinine; Day 5; n=9, 9 | 79.57 (17.196) | 80.33 (11.925)
  Total bilirubin; Baseline; n=18, 18 | 10.56 (3.578) | 10.56 (3.578)
  Total bilirubin; Day 2; n=18, 18 | 11.45 (4.334) | 10.91 (2.952)
  Total bilirubin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Total bilirubin; Day 5; n=9, 9 | 11.49 (1.590) | 11.41 (3.867)
  Direct bilirubin; Baseline; n=18, 18 | 1.96 (0.624) | 1.96 (0.624)
  Direct bilirubin; Day 2; n=18, 18 | 1.91 (0.643) | 1.86 (0.631)
  Direct bilirubin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Direct bilirubin; Day 5; n=9, 9 | 1.86 (0.332) | 1.90 (0.752)
  Urate; Baseline; n=18, 18 | 306.7 (87.16) | 306.7 (87.16)
  Urate; Day 2; n=18, 18 | 283.2 (78.74) | 282.5 (68.93)
  Urate; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Urate; Day 5; n=9, 9 | 281.4 (75.17) | 282.9 (67.35)

36. Secondary Outcome: Absolute Values for Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, Chloride, Phosphate, Blood Urea Nitrogen (BUN), Triglycerides, Cholesterol, Anion Gap, Carbon Dioxide-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: calcium, glucose, potassium, sodium, chloride, phosphate, BUN, triglycerides, cholesterol, anion gap and carbon dioxide.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Millimoles per liter
  Calcium; Baseline; n=18, 18 | 2.327 (0.0451) | 2.327 (0.0451)
  Calcium; Day 2; n=18, 18 | 2.352 (0.0536) | 2.378 (0.0830)
  Calcium; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Calcium; Day 5; n=9, 9 | 2.343 (0.0705) | 2.313 (0.0559)
  Glucose; Baseline; n=18, 18 | 4.987 (0.3833) | 4.987 (0.3833)
  Glucose; Day 2; n=18, 18 | 4.842 (0.3451) | 4.706 (0.2996)
  Glucose; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Glucose; Day 5; n=9, 9 | 4.607 (0.2889) | 4.600 (0.2182)
  Potassium; Baseline; n=18, 18 | 4.00 (0.230) | 4.00 (0.230)
  Potassium; Day 2; n=18, 18 | 4.27 (0.256) | 4.33 (0.379)
  Potassium; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Potassium; Day 5; n=9, 9 | 4.18 (0.228) | 4.13 (0.320)
  Sodium; Baseline; n=18, 18 | 136.9 (2.19) | 136.9 (2.19)
  Sodium; Day 2; n=18, 18 | 138.5 (1.54) | 138.9 (1.75)
  Sodium; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Sodium; Day 5; n=9, 9 | 138.2 (1.48) | 138.8 (1.48)
  Chloride; Baseline; n=18, 18 | 102.3 (1.64) | 102.3 (1.64)
  Chloride; Day 2; n=18, 18 | 102.5 (1.69) | 102.9 (1.66)
  Chloride; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Chloride; Day 5; n=9, 9 | 101.9 (1.76) | 101.8 (1.56)
  Phosphate; Baseline; n=18, 18 | 1.121 (0.1289) | 1.121 (0.1289)
  Phosphate; Day 2; n=18, 18 | 1.197 (0.1058) | 1.197 (0.1365)
  Phosphate; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Phosphate; Day 5; n=9, 9 | 1.173 (0.1413) | 1.234 (0.0963)
  BUN; Baseline; n=18, 18 | 3.728 (1.0672) | 3.728 (1.0672)
  BUN; Day 2; n=18, 18 | 4.747 (0.8949) | 4.654 (0.8997)
  BUN; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  BUN; Day 5; n=9, 9 | 5.053 (0.9143) | 4.729 (0.7928)
  Triglycerides; Baseline; n=18, 18 | 1.026 (0.6064) | 1.026 (0.6064)
  Triglycerides; Day 2; n=18, 18 | 1.127 (0.3973) | 1.036 (0.3982)
  Triglycerides; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Triglycerides; Day 5; n=9, 9 | 1.029 (0.3389) | 0.904 (0.2605)
  Cholesterol; Baseline; n=18, 18 | 4.549 (0.9656) | 4.549 (0.9656)
  Cholesterol; Day 2; n=18, 18 | 4.544 (0.8853) | 4.632 (0.9164)
  Cholesterol; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Cholesterol; Day 5; n=9, 9 | 4.519 (0.6212) | 4.330 (1.1611)
  Anion gap; Baseline; n=18, 18 | 9.5 (1.76) | 9.5 (1.76)
  Anion gap; Day 2; n=18, 18 | 10.1 (1.28) | 10.0 (1.08)
  Anion gap; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Anion gap; Day 5; n=9, 9 | 10.7 (0.87) | 10.1 (0.93)
  Carbon dioxide; Baseline; n=18, 18 | 29.1 (2.00) | 29.1 (2.00)
  Carbon dioxide; Day 2; n=18, 18 | 30.1 (1.86) | 30.2 (1.58)
  Carbon dioxide; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Carbon dioxide; Day 5; n=9, 9 | 29.9 (1.36) | 31.0 (1.87)

37. Secondary Outcome: Absolute Values for Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), Gamma-glutamyl Transferase (GGT), Creatine Kinase (CK), Lactate Dehydrogenase (LDH)-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: ALT, ALP, AST, GGT, CK and LDH.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
International units per liter
  ALT; Baseline; n=18, 18 | 22.1 (12.44) | 22.1 (12.44)
  ALT; Day 2; n=18, 18 | 21.8 (13.38) | 18.4 (9.28)
  ALT; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  ALT; Day 5; n=9, 9 | 20.6 (14.51) | 19.6 (7.07)
  ALP; Baseline; n=18, 18 | 54.6 (11.32) | 54.6 (11.32)
  ALP; Day 2; n=18, 18 | 52.1 (11.59) | 52.1 (10.96)
  ALP; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  ALP; Day 5; n=9, 9 | 55.2 (12.34) | 50.3 (5.87)
  AST; Baseline; n=18, 18 | 21.7 (8.39) | 21.7 (8.39)
  AST; Day 2; n=18, 18 | 19.1 (6.65) | 17.6 (4.94)
  AST; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  AST; Day 5; n=9, 9 | 19.0 (4.30) | 17.0 (3.71)
  GGT; Baseline; n=18, 18 | 19.3 (11.26) | 19.3 (11.26)
  GGT; Day 2; n=18, 18 | 18.1 (11.18) | 18.9 (11.60)
  GGT; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  GGT; Day 5; n=9, 9 | 19.2 (13.07) | 15.8 (6.85)
  CK; Baseline; n=18, 18 | 126.9 (62.61) | 126.9 (62.61)
  CK; Day 2; n=18, 18 | 87.4 (40.30) | 92.2 (44.64)
  CK; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  CK; Day 5; n=9, 9 | 86.0 (35.27) | 98.3 (50.21)
  LDH; Baseline; n=18, 18 | 136.4 (20.82) | 136.4 (20.82)
  LDH; Day 2; n=18, 18 | 117.7 (21.06) | 120.4 (21.17)
  LDH; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  LDH; Day 5; n=9, 9 | 122.0 (20.91) | 123.6 (18.53)

38. Secondary Outcome: Absolute Values for Chemistry Parameters: Albumin, Globulin and Protein-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: albumin, globulin and protein.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Grams per liter
  Albumin; Baseline; n=18, 18 | 43.7 (2.52) | 43.7 (2.52)
  Albumin; Day 2; n=18, 18 | 43.8 (2.53) | 44.4 (2.96)
  Albumin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Albumin; Day 5; n=9, 9 | 45.1 (2.85) | 44.2 (2.82)
  Globulin; Baseline; n=18, 18 | 27.5 (3.84) | 27.5 (3.84)
  Globulin; Day 2; n=18, 18 | 26.9 (4.58) | 27.8 (4.35)
  Globulin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Globulin; Day 5; n=9, 9 | 26.2 (4.58) | 28.0 (4.97)
  Protein; Baseline; n=18, 18 | 71.2 (3.19) | 71.2 (3.19)
  Protein; Day 2; n=18, 18 | 70.7 (5.07) | 72.2 (5.43)
  Protein; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Protein; Day 5; n=9, 9 | 71.3 (6.42) | 72.2 (4.74)

39. Secondary Outcome: Absolute Values for Chemistry Parameters: Amylase and Lipase-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: amylase and lipase.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Units per liter
  Amylase; Baseline; n=18, 18 | 43.3 (14.96) | 43.3 (14.96)
  Amylase; Day 2; n=18, 18 | 46.7 (18.11) | 47.7 (21.31)
  Amylase; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Amylase; Day 5; n=9, 9 | 44.3 (15.86) | 47.6 (22.94)
  Lipase; Baseline; n=18, 18 | 24.0 (11.24) | 24.0 (11.24)
  Lipase; Day 2; n=18, 18 | 26.7 (14.32) | 26.2 (14.26)
  Lipase; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Lipase; Day 5; n=9, 9 | 28.9 (14.98) | 24.7 (12.66)

40. Secondary Outcome: Absolute Values for Chemistry Parameters: Creatinine, Total Bilirubin, Direct Bilirubin and Urate-Part 2
Description: as for outcome 35
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Micromoles per liter
  Creatinine; Baseline; n=20, 19, 21 | 74.00 (13.855) | 74.00 (13.855) | 74.00 (13.855)
  Creatinine; Day 2; n=20, 19, 21 | 81.95 (14.968) | 83.34 (11.078) | 80.18 (13.533)
  Creatinine; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Creatinine; Day 5; n=7, 5, 7 | 91.69 (7.992) | 76.04 (14.435) | 83.71 (15.520)
  Total bilirubin; Baseline; n=20, 19, 21 | 9.05 (3.070) | 9.05 (3.070) | 9.05 (3.070)
  Total bilirubin; Day 2; n=20, 19, 21 | 11.49 (4.185) | 11.88 (4.544) | 11.11 (3.517)
  Total bilirubin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Total bilirubin; Day 5; n=7, 5, 7 | 13.34 (4.999) | 14.30 (7.174) | 10.46 (1.397)
  Direct bilirubin; Baseline; n=20, 19, 21 | 1.89 (0.660) | 1.89 (0.660) | 1.89 (0.660)
  Direct bilirubin; Day 2; n=20, 19, 21 | 2.12 (0.747) | 2.17 (0.732) | 2.07 (0.656)
  Direct bilirubin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Direct bilirubin; Day 5; n=7, 5, 7 | 2.29 (0.760) | 2.38 (0.996) | 1.87 (0.431)
  Urate; Baseline; n=20, 19, 21 | 289.2 (73.13) | 289.2 (73.13) | 289.2 (73.13)
  Urate; Day 2; n=20, 19, 21 | 277.7 (72.39) | 299.4 (68.62) | 275.4 (77.75)
  Urate; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Urate; Day 5; n=7, 5, 7 | 286.3 (48.83) | 291.2 (96.66) | 313.6 (79.74)

41. Secondary Outcome: Absolute Values for Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, Chloride, Phosphate, BUN, Triglycerides, Cholesterol, Anion Gap, Carbon Dioxide-Part 2
Description: as for outcome 36
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Millimoles per liter
  Calcium; Baseline; n=20, 19, 21 | 2.312 (0.0973) | 2.312 (0.0973) | 2.312 (0.0973)
  Calcium; Day 2; n=20, 19, 21 | 2.408 (0.0670) | 2.369 (0.0671) | 2.390 (0.0695)
  Calcium; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Calcium; Day 5; n=7, 5, 7 | 2.446 (0.0500) | 2.324 (0.0439) | 2.367 (0.0640)
  Glucose; Baseline; n=20, 19, 21 | 4.745 (0.3160) | 4.745 (0.3160) | 4.745 (0.3160)
  Glucose; Day 2; n=20, 19, 21 | 4.716 (0.2093) | 4.861 (0.2250) | 4.775 (0.2039)
  Glucose; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Glucose; Day 5; n=7, 5, 7 | 4.574 (0.3675) | 4.608 (0.3518) | 4.926 (0.2224)
  Potassium; Baseline; n=20, 19, 21 | 4.16 (0.225) | 4.16 (0.225) | 4.16 (0.225)
  Potassium; Day 2; n=20, 19, 21 | 4.26 (0.244) | 4.17 (0.281) | 4.14 (0.240)
  Potassium; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Potassium; Day 5; n=7, 5, 7 | 3.84 (0.251) | 3.94 (0.230) | 4.17 (0.236)
  Sodium; Baseline; n=20, 19, 21 | 138.4 (1.56) | 138.4 (1.56) | 138.4 (1.56)
  Sodium; Day 2; n=20, 19, 21 | 137.9 (2.00) | 137.9 (2.58) | 137.4 (1.24)
  Sodium; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Sodium; Day 5; n=7, 5, 7 | 137.3 (1.11) | 136.2 (2.59) | 136.3 (1.89)
  Chloride; Baseline; n=20, 19, 21 | 102.4 (1.72) | 102.4 (1.72) | 102.4 (1.72)
  Chloride; Day 2; n=20, 19, 21 | 102.0 (1.81) | 102.2 (2.06) | 102.0 (2.09)
  Chloride; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Chloride; Day 5; n=7, 5, 7 | 100.3 (1.38) | 101.8 (2.28) | 100.4 (2.37)
  Phosphate; Baseline; n=20, 19, 21 | 1.100 (0.1813) | 1.100 (0.1813) | 1.100 (0.1813)
  Phosphate; Day 2; n=20, 19, 21 | 1.191 (0.1827) | 1.177 (0.1535) | 1.176 (0.1730)
  Phosphate; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Phosphate; Day 5; n=7, 5, 7 | 1.297 (0.1577) | 1.158 (0.2958) | 1.117 (0.1612)
  BUN; Baseline; n=20, 19, 21 | 4.190 (0.9187) | 4.190 (0.9187) | 4.190 (0.9187)
  BUN; Day 2; n=20, 19, 21 | 4.526 (0.7144) | 4.531 (0.8261) | 4.403 (0.8736)
  BUN; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  BUN; Day 5; n=7, 5, 7 | 4.921 (0.9744) | 4.768 (0.4098) | 5.050 (1.2701)
  Triglycerides; Baseline; n=20, 19, 21 | 0.828 (0.3752) | 0.828 (0.3752) | 0.828 (0.3752)
  Triglycerides; Day 2; n=20, 19, 21 | 0.957 (0.3872) | 0.994 (0.3875) | 0.890 (0.4024)
  Triglycerides; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Triglycerides; Day 5; n=7, 5, 7 | 0.894 (0.3072) | 0.774 (0.2790) | 1.363 (0.6417)
  Cholesterol; Baseline; n=20, 19, 21 | 4.533 (0.8776) | 4.533 (0.8776) | 4.533 (0.8776)
  Cholesterol; Day 2; n=20, 19, 21 | 4.652 (0.7742) | 4.639 (0.9975) | 4.610 (0.8031)
  Cholesterol; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Cholesterol; Day 5; n=7, 5, 7 | 4.520 (0.5269) | 3.962 (0.8236) | 4.454 (0.8948)
  Anion gap; Baseline; n=20, 19, 21 | 11.3 (1.53) | 11.3 (1.53) | 11.3 (1.53)
  Anion gap; Day 2; n=20, 19, 21 | 10.6 (1.15) | 10.4 (1.17) | 10.8 (1.54)
  Anion gap; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Anion gap; Day 5; n=7, 5, 7 | 11.7 (2.43) | 10.8 (0.84) | 11.9 (1.68)
  Carbon dioxide; Baseline; n=20, 19, 21 | 28.7 (2.00) | 28.7 (2.00) | 28.7 (2.00)
  Carbon dioxide; Day 2; n=20, 19, 21 | 29.6 (1.67) | 29.5 (1.78) | 28.6 (2.20)
  Carbon dioxide; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Carbon dioxide; Day 5; n=7, 5, 7 | 29.3 (1.50) | 27.6 (2.19) | 28.1 (1.57)

42. Secondary Outcome: Absolute Values for Chemistry Parameters: ALT, ALP, AST, GGT, CK, LDH-Part 2
Description: as for outcome 37
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
International units per liter
  ALT; Baseline; n=20, 19, 21 | 19.0 (11.01) | 19.0 (11.01) | 19.0 (11.01)
  ALT; Day 2; n=20, 19, 21 | 14.4 (6.06) | 17.3 (9.49) | 16.8 (9.20)
  ALT; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  ALT; Day 5; n=7, 5, 7 | 16.7 (8.04) | 11.0 (2.74) | 22.7 (14.36)
  ALP; Baseline; n=20, 19, 21 | 50.4 (16.47) | 50.4 (16.47) | 50.4 (16.47)
  ALP; Day 2; n=20, 19, 21 | 56.5 (17.52) | 57.4 (17.03) | 56.7 (18.33)
  ALP; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  ALP; Day 5; n=7, 5, 7 | 49.6 (22.40) | 56.4 (9.58) | 55.0 (13.69)
  AST; Baseline; n=20, 19, 21 | 18.0 (6.01) | 18.0 (6.01) | 18.0 (6.01)
  AST; Day 2; n=20, 19, 21 | 14.9 (3.01) | 15.8 (4.29) | 16.0 (4.11)
  AST; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  AST; Day 5; n=7, 5, 7 | 16.7 (4.42) | 14.0 (2.12) | 16.6 (3.78)
  GGT; Baseline; n=20, 19, 21 | 17.1 (5.80) | 17.1 (5.80) | 17.1 (5.80)
  GGT; Day 2; n=20, 19, 21 | 16.5 (5.56) | 17.4 (6.15) | 17.3 (7.67)
  GGT; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  GGT; Day 5; n=7, 5, 7 | 14.9 (3.72) | 14.8 (0.45) | 21.6 (13.31)
  CK; Baseline; n=20, 19, 21 | 118.8 (79.80) | 118.8 (79.80) | 118.8 (79.80)
  CK; Day 2; n=20, 19, 21 | 106.2 (80.82) | 114.9 (101.61) | 106.2 (81.94)
  CK; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  CK; Day 5; n=7, 5, 7 | 135.7 (108.77) | 136.4 (109.71) | 145.4 (170.90)
  LDH; Baseline; n=20, 19, 21 | 133.6 (19.21) | 133.6 (19.21) | 133.6 (19.21)
  LDH; Day 2; n=20, 19, 21 | 121.1 (17.48) | 121.5 (21.60) | 122.1 (18.56)
  LDH; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  LDH; Day 5; n=7, 5, 7 | 118.4 (16.63) | 110.0 (12.29) | 126.0 (22.84)

43. Secondary Outcome: Absolute Values for Chemistry Parameters: Albumin, Globulin and Protein-Part 2
Description: as for outcome 38
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Grams per liter
  Albumin; Baseline; n=20, 19, 21 | 43.8 (2.90) | 43.8 (2.90) | 43.8 (2.90)
  Albumin; Day 2; n=20, 19, 21 | 45.6 (2.68) | 45.4 (2.27) | 45.7 (2.99)
  Albumin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Albumin; Day 5; n=7, 5, 7 | 48.0 (2.58) | 43.4 (2.07) | 45.1 (2.97)
  Globulin; Baseline; n=20, 19, 21 | 26.5 (3.19) | 26.5 (3.19) | 26.5 (3.19)
  Globulin; Day 2; n=20, 19, 21 | 26.6 (3.33) | 26.0 (3.43) | 26.4 (3.43)
  Globulin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Globulin; Day 5; n=7, 5, 7 | 23.6 (1.51) | 28.2 (2.49) | 26.7 (1.25)
  Protein; Baseline; n=20, 19, 21 | 70.3 (4.23) | 70.3 (4.23) | 70.3 (4.23)
  Protein; Day 2; n=20, 19, 21 | 72.2 (3.56) | 71.4 (3.20) | 72.1 (4.31)
  Protein; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Protein; Day 5; n=7, 5, 7 | 71.6 (3.15) | 71.6 (2.07) | 71.9 (2.85)

44. Secondary Outcome: Absolute Values for Chemistry Parameters: Amylase and Lipase-Part 2
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: amylase and lipase.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Units per liter
  Amylase; Baseline; n=20, 19, 21 | 49.3 (16.33) | 49.3 (16.33) | 49.3 (16.33)
  Amylase; Day 2; n=20, 19, 21 | 48.3 (15.91) | 49.4 (18.86) | 50.1 (18.22)
  Amylase; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Amylase; Day 5; n=7, 5, 7 | 49.6 (22.33) | 48.8 (8.53) | 43.6 (14.89)
  Lipase; Baseline; n=20, 19, 21 | 23.8 (17.88) | 23.8 (17.88) | 23.8 (17.88)
  Lipase; Day 2; n=20, 19, 21 | 20.4 (10.04) | 22.2 (12.81) | 24.1 (11.45)
  Lipase; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Lipase; Day 5; n=7, 5, 7 | 21.9 (9.39) | 17.6 (8.23) | 24.1 (13.26)

45. Secondary Outcome: Change From Baseline Chemistry Parameters: Creatinine, Total Bilirubin, Direct Bilirubin and Urate-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: creatinine, total bilirubin, direct bilirubin and urate. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Micromoles per liter
  Creatinine; Day 2; n=18, 18 | 2.19 (4.721) | 1.43 (6.188)
  Creatinine; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Creatinine; Day 5; n=9, 9 | 3.64 (3.780) | -1.10 (5.169)
  Total bilirubin; Day 2; n=18, 18 | 0.89 (2.659) | 0.36 (2.632)
  Total bilirubin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Total bilirubin; Day 5; n=9, 9 | 0.59 (3.297) | 1.20 (2.513)
  Direct bilirubin; Day 2; n=18, 18 | -0.05 (0.399) | -0.10 (0.387)
  Direct bilirubin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Direct bilirubin; Day 5; n=9, 9 | -0.12 (0.526) | -0.04 (0.361)
  Urate; Day 2; n=18, 18 | -23.5 (46.62) | -24.2 (43.16)
  Urate; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Urate; Day 5; n=9, 9 | -29.8 (46.45) | -19.3 (36.96)

46. Secondary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, Chloride, Phosphate, BUN, Triglycerides, Cholesterol, Anion Gap, Carbon Dioxide-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: calcium, glucose, potassium, sodium, chloride, phosphate, BUN, triglycerides, cholesterol, anion gap and carbon dioxide. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Millimoles per liter
  Calcium; Day 2; n=18, 18 | 0.025 (0.0534) | 0.051 (0.0828)
  Calcium; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Calcium; Day 5; n=9, 9 | 0.019 (0.0762) | -0.016 (0.0548)
  Glucose; Day 2; n=18, 18 | -0.145 (0.3134) | -0.281 (0.4796)
  Glucose; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Glucose; Day 5; n=9, 9 | -0.252 (0.4474) | -0.514 (0.3475)
  Potassium; Day 2; n=18, 18 | 0.27 (0.278) | 0.33 (0.331)
  Potassium; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Potassium; Day 5; n=9, 9 | 0.30 (0.296) | 0.01 (0.247)
  Sodium; Day 2; n=18, 18 | 1.6 (2.30) | 2.0 (2.28)
  Sodium; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Sodium; Day 5; n=9, 9 | 1.8 (2.77) | 1.4 (1.33)
  Chloride; Day 2; n=18, 18 | 0.2 (2.05) | 0.7 (2.22)
  Chloride; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Chloride; Day 5; n=9, 9 | -0.2 (2.33) | -0.7 (1.73)
  Phosphate; Day 2; n=18, 18 | 0.077 (0.1177) | 0.077 (0.1223)
  Phosphate; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Phosphate; Day 5; n=9, 9 | 0.077 (0.1331) | 0.090 (0.1282)
  BUN; Day 2; n=18, 18 | 1.019 (0.9553) | 0.926 (1.0408)
  BUN; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  BUN; Day 5; n=9, 9 | 1.178 (1.0554) | 1.148 (0.6297)
  Triglycerides; Day 2; n=18, 18 | 0.101 (0.4182) | 0.010 (0.4769)
  Triglycerides; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Triglycerides; Day 5; n=9, 9 | 0.102 (0.2870) | -0.221 (0.5382)
  Cholesterol; Day 2; n=18, 18 | -0.005 (0.3983) | 0.082 (0.4981)
  Cholesterol; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Cholesterol; Day 5; n=9, 9 | -0.148 (0.4463) | -0.102 (0.6612)
  Anion gap; Day 2; n=18, 18 | 0.6 (2.03) | 0.5 (1.95)
  Anion gap; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Anion gap; Day 5; n=9, 9 | 0.8 (2.64) | 1.0 (1.22)
  Carbon dioxide; Day 2; n=18, 18 | 0.9 (2.60) | 1.1 (2.10)
  Carbon dioxide; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Carbon dioxide; Day 5; n=9, 9 | 1.4 (2.60) | 1.2 (1.56)

47. Secondary Outcome: Change From Baseline in Chemistry Parameters: ALT, ALP, AST, GGT, CK, LDH-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: ALT, ALP, AST, GGT, CK and LDH. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
International units per liter
  ALT; Day 2; n=18, 18 | -0.2 (5.34) | -3.6 (8.39)
  ALT; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  ALT; Day 5; n=9, 9 | 1.3 (7.87) | -5.3 (12.32)
  ALP; Day 2; n=18, 18 | -2.4 (5.25) | -2.5 (4.74)
  ALP; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  ALP; Day 5; n=9, 9 | -1.7 (7.40) | -1.9 (3.37)
  AST; Day 2; n=18, 18 | -2.6 (4.68) | -4.2 (6.57)
  AST; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  AST; Day 5; n=9, 9 | -1.4 (3.84) | -6.0 (8.70)
  GGT; Day 2; n=18, 18 | -1.2 (1.93) | -0.4 (2.94)
  GGT; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  GGT; Day 5; n=9, 9 | -2.1 (2.47) | -1.6 (3.88)
  CK; Day 2; n=18, 18 | -39.6 (39.29) | -34.8 (53.99)
  CK; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  CK; Day 5; n=9, 9 | -23.3 (28.33) | -46.2 (76.08)
  LDH; Day 2; n=18, 18 | -18.7 (11.00) | -16.0 (11.86)
  LDH; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  LDH; Day 5; n=9, 9 | -13.9 (16.12) | -13.4 (16.13)

48. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin, Globulin and Protein-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: albumin, globulin and protein. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Grams per liter
  Albumin; Day 2; n=18, 18 | 0.1 (2.80) | 0.7 (3.04)
  Albumin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Albumin; Day 5; n=9, 9 | 0.9 (3.37) | 1.0 (3.00)
  Globulin; Day 2; n=18, 18 | -0.6 (2.50) | 0.3 (2.37)
  Globulin; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Globulin; Day 5; n=9, 9 | -0.7 (2.78) | -0.1 (1.76)
  Protein; Day 2; n=18, 18 | -0.5 (4.82) | 1.0 (4.79)
  Protein; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Protein; Day 5; n=9, 9 | 0.2 (5.93) | 0.9 (4.54)

49. Secondary Outcome: Change From Baseline in Chemistry Parameters: Amylase and Lipase-Part 1
Description: Blood samples were collected for the assessment of following clinical chemistry parameters: amylase and lipase. Baseline value was the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Units per liter
  Amylase; Day 2; n=18, 18 | 3.3 (5.66) | 4.3 (8.75)
  Amylase; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Amylase; Day 5; n=9, 9 | 1.0 (6.52) | 4.2 (6.22)
  Lipase; Day 2; n=18, 18 | 2.7 (8.27) | 2.2 (5.15)
  Lipase; Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Lipase; Day 5; n=9, 9 | 4.0 (6.56) | 1.6 (3.28)

50. Secondary Outcome: Change From Baseline in Chemistry Parameters: Creatinine, Total Bilirubin, Direct Bilirubin and Urate-Part 2
Description: as for outcome 45
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Micromoles per liter
  Creatinine; Day 2; n=20, 19, 21 | 7.25 (5.306) | 7.41 (4.836) | 6.18 (4.833)
  Creatinine; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Creatinine; Day 5; n=7, 5, 7 | 10.10 (5.536) | 8.86 (4.565) | 7.19 (5.827)
  Total bilirubin; Day 2; n=20, 19, 21 | 2.29 (2.650) | 2.47 (3.448) | 2.06 (2.729)
  Total bilirubin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Total bilirubin; Day 5; n=7, 5, 7 | 3.89 (3.133) | 4.04 (4.689) | 1.69 (1.791)
  Direct bilirubin; Day 2; n=20, 19, 21 | 0.21 (0.524) | 0.22 (0.550) | 0.18 (0.494)
  Direct bilirubin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Direct bilirubin; Day 5; n=7, 5, 7 | 0.31 (0.495) | 0.16 (0.611) | 0.11 (0.389)
  Urate; Day 2; n=20, 19, 21 | -16.5 (31.57) | -0.5 (29.49) | -13.8 (32.92)
  Urate; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Urate; Day 5; n=7, 5, 7 | -6.7 (29.86) | -4.0 (34.62) | 3.3 (27.67)

51. Secondary Outcome: Change From Baseline in Chemistry Parameters: Calcium, Glucose, Potassium, Sodium, Chloride, Phosphate, BUN, Triglycerides, Cholesterol, Anion Gap, Carbon Dioxide-Part 2
Description: as for outcome 46
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Millimoles per liter
  Calcium; Day 2; n=20, 19, 21 | 0.098 (0.0777) | 0.063 (0.0930) | 0.078 (0.0590)
  Calcium; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Calcium; Day 5; n=7, 5, 7 | 0.097 (0.0663) | 0.068 (0.0867) | 0.067 (0.0702)
  Glucose; Day 2; n=20, 19, 21 | -0.036 (0.2823) | 0.087 (0.2938) | 0.030 (0.2588)
  Glucose; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Glucose; Day 5; n=7, 5, 7 | -0.207 (0.3073) | -0.100 (0.2547) | 0.113 (0.3935)
  Potassium; Day 2; n=20, 19, 21 | 0.08 (0.249) | -0.01 (0.273) | -0.02 (0.270)
  Potassium; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Potassium; Day 5; n=7, 5, 7 | -0.26 (0.270) | -0.32 (0.377) | -0.04 (0.282)
  Sodium; Day 2; n=20, 19, 21 | -0.5 (2.06) | -0.5 (2.59) | -1.0 (2.00)
  Sodium; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Sodium; Day 5; n=7, 5, 7 | -1.9 (0.69) | -2.0 (1.41) | -1.4 (3.10)
  Chloride; Day 2; n=20, 19, 21 | -0.5 (1.67) | -0.2 (1.78) | -0.3 (2.29)
  Chloride; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Chloride; Day 5; n=7, 5, 7 | -1.9 (0.90) | -2.2 (1.10) | -1.0 (2.89)
  Phosphate; Day 2; n=20, 19, 21 | 0.087 (0.0836) | 0.065 (0.0973) | 0.076 (0.0815)
  Phosphate; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Phosphate; Day 5; n=7, 5, 7 | 0.060 (0.0856) | 0.124 (0.0953) | 0.074 (0.0820)
  BUN; Day 2; n=20, 19, 21 | 0.307 (0.8732) | 0.257 (0.9884) | 0.213 (0.9258)
  BUN; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  BUN; Day 5; n=7, 5, 7 | 0.783 (1.1942) | 0.684 (0.7695) | 0.506 (0.9007)
  Triglycerides; Day 2; n=20, 19, 21 | 0.115 (0.2130) | 0.127 (0.2750) | 0.062 (0.2884)
  Triglycerides; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Triglycerides; Day 5; n=7, 5, 7 | 0.021 (0.2874) | 0.226 (0.1254) | 0.273 (0.5007)
  Cholesterol; Day 2; n=20, 19, 21 | 0.103 (0.4625) | 0.078 (0.5175) | 0.077 (0.4478)
  Cholesterol; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Cholesterol; Day 5; n=7, 5, 7 | -0.033 (0.5333) | -0.286 (0.3791) | -0.339 (0.3855)
  Anion gap; Day 2; n=20, 19, 21 | -0.8 (1.41) | -0.9 (2.13) | -0.5 (1.66)
  Anion gap; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Anion gap; Day 5; n=7, 5, 7 | 1.0 (1.73) | 0.4 (1.67) | -0.7 (1.98)
  Carbon dioxide; Day 2; n=20, 19, 21 | 0.9 (1.59) | 0.8 (1.18) | -0.1 (2.10)
  Carbon dioxide; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Carbon dioxide; Day 5; n=7, 5, 7 | -1.0 (2.00) | -0.4 (2.30) | 0.4 (1.81)

52. Secondary Outcome: Change From Baseline in Chemistry Parameters: ALT, ALP, AST, GGT, CK, LDH-Part 2
Description: as for outcome 47
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
International units per liter
  ALT; Day 2; n=20, 19, 21 | -4.9 (8.61) | -2.5 (4.06) | -2.2 (8.48)
  ALT; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  ALT; Day 5; n=7, 5, 7 | -9.7 (13.03) | -3.4 (4.39) | 5.7 (9.23)
  ALP; Day 2; n=20, 19, 21 | 6.1 (5.61) | 5.9 (5.91) | 6.3 (6.21)
  ALP; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  ALP; Day 5; n=7, 5, 7 | 3.9 (6.69) | 2.2 (6.22) | -0.4 (6.50)
  AST; Day 2; n=20, 19, 21 | -3.3 (5.18) | -2.6 (4.40) | -2.0 (4.88)
  AST; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  AST; Day 5; n=7, 5, 7 | -5.1 (6.26) | -2.8 (4.66) | 0.6 (3.36)
  GGT; Day 2; n=20, 19, 21 | -1.1 (2.65) | -0.4 (1.80) | 0.2 (3.09)
  GGT; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  GGT; Day 5; n=7, 5, 7 | -2.4 (3.31) | -1.4 (2.70) | 2.1 (5.73)
  CK; Day 2; n=20, 19, 21 | -15.4 (27.15) | -10.7 (40.57) | -12.6 (31.50)
  CK; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  CK; Day 5; n=7, 5, 7 | 1.1 (78.79) | 9.4 (92.62) | 29.9 (152.85)
  LDH; Day 2; n=20, 19, 21 | -12.2 (10.28) | -12.4 (12.05) | -11.5 (11.97)
  LDH; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  LDH; Day 5; n=7, 5, 7 | -17.3 (14.95) | -17.8 (3.27) | -10.4 (15.05)

53. Secondary Outcome: Change From Baseline in Chemistry Parameters: Albumin, Globulin and Protein-Part 2
Description: as for outcome 48
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Grams per liter
  Albumin; Day 2; n=20, 19, 21 | 2.0 (1.85) | 1.8 (2.57) | 1.9 (1.95)
  Albumin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Albumin; Day 5; n=7, 5, 7 | 3.4 (1.40) | 1.8 (0.84) | 1.1 (1.46)
  Globulin; Day 2; n=20, 19, 21 | 0.2 (1.79) | -0.1 (2.26) | -0.1 (1.76)
  Globulin; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Globulin; Day 5; n=7, 5, 7 | 0.1 (1.86) | 0.1 (3.39) | -1.3 (1.80)
  Protein; Day 2; n=20, 19, 21 | 2.1 (3.01) | 1.7 (4.28) | 1.8 (3.01)
  Protein; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Protein; Day 5; n=7, 5, 7 | 3.6 (2.23) | 2.8 (4.09) | -0.1 (3.02)

54. Secondary Outcome: Change From Baseline in Chemistry Parameters: Amylase and Lipase-Part 2
Description: as for outcome 49
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Units per liter
  Amylase; Day 2; n=20, 19, 21 | 0.7 (5.68) | 1.8 (8.70) | 0.8 (8.27)
  Amylase; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Amylase; Day 5; n=7, 5, 7 | 4.4 (4.86) | -1.8 (10.16) | -4.4 (8.26)
  Lipase; Day 2; n=20, 19, 21 | -2.6 (15.99) | -1.4 (13.01) | 0.3 (17.39)
  Lipase; Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Lipase; Day 5; n=7, 5, 7 | 6.3 (7.54) | -3.0 (14.27) | -9.6 (24.84)

55. Secondary Outcome: Absolute Values for Urine Parameter: Specific Gravity-Part 1
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine, indicated as ratio of urine density to water density.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Ratio
  Baseline; n=18, 18 | 1.0120 (0.00915) | 1.0120 (0.00915)
  Day 2; n=18, 18 | 1.0152 (0.00685) | 1.0158 (0.00584)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 1.0201 (0.00664) | 1.0161 (0.00434)

56. Secondary Outcome: Absolute Values for Urine Parameter: Urobilinogen-Part 1
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Micromoles per liter
  Baseline; n=18, 18 | 4.1384 (3.19235) | 4.1384 (3.19235)
  Day 2; n=18, 18 | 3.3860 (0.00000) | 4.1384 (3.19235)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 3.3860 (0.00000) | 3.3860 (0.00000)

57. Secondary Outcome: Absolute Values for Urine Parameter: Potential of Hydrogen (pH)-Part 1
Description: Urine samples were collected at indicated time points for the assessment of urine pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0).
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
pH
  Baseline; n=18, 18 | 6.03 (0.696) | 6.03 (0.696)
  Day 2; n=18, 18 | 6.14 (0.682) | 6.25 (0.600)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 5.72 (0.441) | 5.89 (0.697)

58. Secondary Outcome: Absolute Values for Urine Parameter: Specific Gravity-Part 2
Description: as for outcome 55
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Ratio
  Baseline; n=20, 19, 21 | 1.0080 (0.00735) | 1.0080 (0.00735) | 1.0080 (0.00735)
  Day 2; n=20, 19, 21 | 1.0166 (0.00675) | 1.0151 (0.00552) | 1.0163 (0.00419)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 1.0180 (0.00632) | 1.0248 (0.00526) | 1.0171 (0.00999)

59. Secondary Outcome: Absolute Values for Urine Parameter: Urobilinogen-Part 2
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Micromoles per liter
  Baseline; n=20, 19, 21 | 4.6759 (4.03794) | 4.6759 (4.03794) | 4.6759 (4.03794)
  Day 2; n=20, 19, 21 | 4.0632 (3.02853) | 3.3860 (0.00000) | 3.3860 (0.00000)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 3.3860 (0.00000) | 6.0948 (6.05706) | 5.3209 (5.11915)

60. Secondary Outcome: Absolute Values for Urine Parameter: pH-Part 2
Description: as for outcome 57
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
pH
  Baseline; n=20, 19, 21 | 6.36 (0.727) | 6.36 (0.727) | 6.36 (0.727)
  Day 2; n=20, 19, 21 | 6.15 (0.690) | 6.08 (0.584) | 6.10 (0.718)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 5.86 (0.627) | 5.60 (0.418) | 6.21 (0.393)

61. Secondary Outcome: Change From Baseline in Urine Parameter: Specific Gravity-Part 1
Description: Urine samples were collected at indicated time points for the assessment of specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine, indicated as ratio of urine density to water density. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Ratio
  Day 2; n=18, 18 | 0.0032 (0.01242) | 0.0038 (0.01043)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 0.0088 (0.01210) | 0.0034 (0.01180)

62. Secondary Outcome: Change From Baseline in Urine Parameter: Urobilinogen-Part 1
Description: Urine samples were collected at indicated time points for the assessment of urine urobilinogen. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Micromoles per liter
  Day 2; n=18, 18 | -0.7524 (3.19235) | 0.0000 (4.64555)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | 0.0000 (0.00000) | -1.5049 (4.51467)

63. Secondary Outcome: Change From Baseline in Urine Parameter: pH-Part 1
Description: Urine samples were collected at indicated time points for the assessment of urine pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits, before the first dose of study drug administration. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
pH
  Day 2; n=18, 18 | 0.11 (1.008) | 0.22 (0.974)
  Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  Day 5; n=9, 9 | -0.17 (0.559) | -0.28 (1.121)

64. Secondary Outcome: Change From Baseline in Urine Parameter: Specific Gravity-Part 2
Description: as for outcome 61
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Ratio
  Day 2; n=20, 19, 21 | 0.0084 (0.00942) | 0.0066 (0.00718) | 0.0083 (0.00728)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 0.0109 (0.00825) | 0.0140 (0.01142) | 0.0091 (0.00956)

65. Secondary Outcome: Change From Baseline in Urine Parameter: Urobilinogen-Part 2
Description: as for outcome 62
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Micromoles per liter
  Day 2; n=20, 19, 21 | -0.6772 (5.33680) | -1.4275 (4.27045) | -1.2899 (4.07394)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | 0.0000 (0.00000) | -2.7088 (6.05706) | 1.9349 (5.11915)

66. Secondary Outcome: Change From Baseline in Urine Parameter: pH-Part 2
Description: as for outcome 63
Time Frame: Baseline (Day -1), Day 2 and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
pH
  Day 2; n=20, 19, 21 | -0.18 (0.799) | -0.18 (0.730) | -0.26 (0.664)
  Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  Day 5; n=7, 5, 7 | -0.43 (0.787) | -0.80 (0.837) | 0.07 (0.450)

67. Secondary Outcome: Number of Participants With Abnormal Urine Dipstick Results-Part 1
Description: Urine samples were collected at indicated time points for the assessment of following urine parameters: bilirubin, glucose, ketones, nitrite, leukocyte esterase, occult blood and protein by dipstick method. The dipstick test gives results in a semi-quantitative manner, and results can be read as Trace, 1+, 2+, 3+ indicating proportional concentrations in the urine sample. Only parameters and time points with abnormal results have been presented.
Time Frame: Day 2 and Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Participants
  Leukocyte esterase, Day 2, Trace | 0 | 1
  Leukocyte esterase, Day 2, 1+ | 1 | 0
  Leukocyte esterase, Day 5, Trace | 0 | 1
  Leukocyte esterase, Day 5, 1+ | 0 | 1
  Occult blood, Day 2, Trace | 1 | 1
  Occult blood, Day 2, 1+ | 1 | 0

68. Secondary Outcome: Number of Participants With Abnormal Urine Dipstick Results-Part 2
Description: as for outcome 67
Time Frame: Day 2 and Day 5
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Participants
  Ketones; Day 5; Trace | 1 | 0 | 0
  Ketones; Day 5; 2+ | 0 | 0 | 1
  Leukocyte esterase; Day 2; 1+ | 0 | 0 | 1
  Occult blood; Day 2; Trace | 0 | 0 | 1
  Occult blood; Day 2; 2+ | 1 | 0 | 0
  Occult blood; Day 2; 3+ | 0 | 0 | 2

69. Secondary Outcome: Absolute Values of Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval and QT Interval Corrected by Fridericia's Formula (QTcF)-Part 1
Description: Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. ECGs were obtained using an ECG machine that automatically measured PR, QRS, QT, and QTcF intervals.
Time Frame: Baseline (Day 1, pre-dose), Day 1 (2 hours and 4 hours) and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Milliseconds
  PR interval, Baseline; n=18, 18 | 164.1 (22.81) | 162.3 (20.76)
  PR interval, Day 1 (2 hours); n=18, 18 | 166.3 (21.55) | 158.7 (19.95)
  PR interval, Day 1 (4 hours); n=18, 18 | 160.6 (20.94) | 158.9 (19.19)
  PR interval, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  PR interval, Day 5; n=9, 9 | 161.8 (11.68) | 169.3 (26.14)
  QRS duration, Baseline; n=18, 18 | 93.4 (9.30) | 92.5 (8.09)
  QRS duration, Day 1 (2 hours); n=18, 18 | 91.9 (8.76) | 92.6 (9.00)
  QRS duration, Day 1 (4 hours); n=18, 18 | 94.1 (8.88) | 93.8 (9.90)
  QRS duration, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  QRS duration, Day 5; n=9, 9 | 94.3 (11.65) | 92.4 (8.25)
  QT interval, Baseline; n=18, 18 | 395.1 (14.22) | 394.4 (24.04)
  QT interval, Day 1 (2 hours); n=18, 18 | 383.3 (13.71) | 383.6 (24.11)
  QT interval, Day 1 (4 hours); n=18, 18 | 404.8 (16.36) | 402.0 (27.67)
  QT interval, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  QT interval, Day 5; n=9, 9 | 393.4 (16.38) | 402.7 (18.71)
  QTcF interval, Baseline; n=18, 18 | 399.4 (9.76) | 401.9 (15.01)
  QTcF interval, Day 1 (2 hours); n=18, 18 | 389.5 (12.11) | 392.8 (15.09)
  QTcF interval, Day 1 (4 hours); n=18, 18 | 398.7 (11.13) | 402.6 (19.46)
  QTcF interval, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  QTcF interval, Day 5; n=9, 9 | 400.8 (13.34) | 399.4 (11.98)

70. Secondary Outcome: Absolute Values of ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF Interval-Part 2
Description: as for outcome 69
Time Frame: Baseline (Day 1, pre-dose), Day 1 (2 hours and 4 hours) and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Milliseconds
  PR interval, Baseline; n=20, 19, 21 | 166.4 (16.48) | 166.2 (15.40) | 166.8 (17.01)
  PR interval, Day 1 (2 hours); n=20, 19, 21 | 163.9 (18.45) | 166.8 (15.23) | 161.7 (16.82)
  PR interval, Day 1 (4 hours); n=20, 19, 21 | 165.2 (17.74) | 165.7 (15.29) | 162.6 (13.99)
  PR interval, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  PR interval, Day 5; n=7, 5, 7 | 173.4 (19.16) | 171.6 (14.57) | 163.1 (12.36)
  QRS duration, Baseline; n=20, 19, 21 | 92.1 (9.76) | 91.7 (9.02) | 90.1 (10.42)
  QRS duration, Day 1 (2 hours); n=20, 19, 21 | 88.9 (9.68) | 92.6 (9.82) | 89.7 (9.86)
  QRS duration, Day 1 (4 hours); n=20, 19, 21 | 91.1 (10.63) | 93.2 (8.45) | 90.3 (8.69)
  QRS duration, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  QRS duration, Day 5; n=7, 5, 7 | 101.1 (7.10) | 85.8 (8.07) | 88.7 (5.28)
  QT interval, Baseline; n=20, 19, 21 | 391.8 (28.22) | 388.5 (24.78) | 389.7 (26.09)
  QT interval, Day 1 (2 hours); n=20, 19, 21 | 379.7 (25.70) | 399.2 (22.43) | 376.2 (22.54)
  QT interval, Day 1 (4 hours); n=20, 19, 21 | 401.0 (25.84) | 406.9 (22.25) | 389.1 (25.95)
  QT interval, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  QT interval, Day 5; n=7, 5, 7 | 401.7 (33.29) | 391.0 (10.27) | 378.9 (25.15)
  QTcF interval, Baseline; n=20, 19, 21 | 395.3 (21.06) | 392.4 (19.45) | 391.9 (21.63)
  QTcF interval, Day 1 (2 hours); n=20, 19, 21 | 384.0 (19.91) | 391.7 (21.77) | 388.3 (18.91)
  QTcF interval, Day 1 (4 hours); n=20, 19, 21 | 396.8 (21.90) | 395.5 (20.75) | 393.3 (20.78)
  QTcF interval, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  QTcF interval, Day 5; n=7, 5, 7 | 391.9 (30.45) | 402.4 (7.70) | 388.1 (22.81)

71. Secondary Outcome: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF Interval-Part 1
Description: Twelve-lead ECGs were performed with the participant in a supine position after a rest of at least 10 minutes. ECGs were obtained using an ECG machine that automatically measured PR, QRS, QT, and QTcF intervals. Baseline is defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Day 1 (2 hours and 4 hours) and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Milliseconds
  PR interval, Day 1 (2 hours); n=18, 18 | 2.2 (8.35) | -3.6 (10.01)
  PR interval, Day 1 (4 hours); n=18, 18 | -3.6 (11.61) | -3.3 (10.85)
  PR interval, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  PR interval, Day 5; n=9, 9 | -0.9 (13.72) | 3.2 (8.35)
  QRS duration, Day 1 (2 hours); n=18, 18 | -1.5 (2.81) | 0.1 (6.06)
  QRS duration, Day 1 (4 hours); n=18, 18 | 0.7 (3.63) | 1.3 (4.92)
  QRS duration, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  QRS duration, Day 5; n=9, 9 | -0.3 (3.74) | 0.8 (3.46)
  QT interval, Day 1 (2 hours); n=18, 18 | -11.8 (10.70) | -10.8 (11.18)
  QT interval, Day 1 (4 hours); n=18, 18 | 9.7 (13.99) | 7.6 (16.85)
  QT interval, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  QT interval, Day 5; n=9, 9 | -1.3 (10.00) | 5.0 (26.51)
  QTcF interval, Day 1 (2 hours); n=18, 18 | -9.9 (6.49) | -9.1 (9.16)
  QTcF interval, Day 1 (4 hours); n=18, 18 | -0.7 (7.71) | 0.7 (9.23)
  QTcF interval, Day 5; n=9, 9: number analyzed (Participants) | 9 | 9
  QTcF interval, Day 5; n=9, 9 | -0.7 (7.19) | 3.9 (7.93)

72. Secondary Outcome: Change From Baseline in ECG Parameters: PR Interval, QRS Duration, QT Interval and QTcF Interval-Part 2
Description: as for outcome 71
Time Frame: Baseline (Day 1, pre-dose), Day 1 (2 hours and 4 hours) and Day 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Milliseconds
  PR interval, Day 1 (2 hours); n=20, 19, 21 | -2.5 (7.02) | 0.7 (7.90) | -5.0 (8.29)
  PR interval, Day 1 (4 hours); n=20, 19, 21 | -1.2 (8.47) | -0.4 (11.52) | -4.2 (6.79)
  PR interval, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  PR interval, Day 5; n=7, 5, 7 | 2.0 (4.08) | 1.6 (11.26) | -2.7 (16.42)
  QRS duration, Day 1 (2 hours); n=20, 19, 21 | -3.2 (3.44) | 0.9 (3.90) | -0.5 (3.03)
  QRS duration, Day 1 (4 hours); n=20, 19, 21 | -1.0 (4.18) | 1.5 (4.45) | 0.2 (4.12)
  QRS duration, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  QRS duration, Day 5; n=7, 5, 7 | 0.4 (3.21) | -0.4 (3.13) | 0.4 (2.88)
  QT interval, Day 1 (2 hours); n=20, 19, 21 | -12.1 (18.05) | 10.6 (12.36) | -13.4 (15.31)
  QT interval, Day 1 (4 hours); n=20, 19, 21 | 9.2 (18.08) | 18.4 (12.90) | -0.6 (14.14)
  QT interval, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  QT interval, Day 5; n=7, 5, 7 | -2.1 (10.67) | -12.4 (13.28) | -2.9 (7.95)
  QTcF interval, Day 1 (2 hours); n=20, 19, 21 | -11.3 (7.04) | -0.6 (7.33) | -3.5 (8.70)
  QTcF interval, Day 1 (4 hours); n=20, 19, 21 | 1.6 (7.50) | 3.1 (7.75) | 1.4 (7.64)
  QTcF interval, Day 5; n=7, 5, 7: number analyzed (Participants) | 7 | 5 | 7
  QTcF interval, Day 5; n=7, 5, 7 | -0.4 (9.34) | -1.4 (3.91) | 1.7 (8.30)

73. Secondary Outcome: Absolute Values for Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)-Part 1
Description: Blood pressure was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Millimeters of mercury
  SBP; Baseline | 118.3 (9.73) | 117.4 (12.26)
  SBP; Day 2 | 113.8 (10.32) | 115.1 (11.94)
  SBP; Day 3 | 113.6 (12.13) | 113.3 (9.71)
  SBP; Day 4 | 112.2 (11.11) | 113.9 (10.57)
  SBP; Day 5 | 112.2 (9.62) | 113.8 (8.91)
  DBP; Baseline | 72.1 (8.35) | 73.4 (8.51)
  DBP; Day 2: number analyzed (Participants) | 9 | 9
  DBP; Day 2 | 70.1 (7.06) | 71.3 (10.56)
  DBP; Day 3 | 70.4 (7.72) | 69.1 (8.46)
  DBP; Day 4 | 70.2 (6.98) | 68.7 (6.77)
  DBP; Day 5 | 70.1 (7.68) | 68.9 (5.76)

74. Secondary Outcome: Absolute Values for Vital Sign: Pulse Rate-Part 1
Description: Pulse rate was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Beats per minute
  Baseline | 65.7 (5.27) | 66.2 (10.00)
  Day 2 | 66.7 (7.02) | 68.4 (8.71)
  Day 3 | 67.4 (7.79) | 68.6 (9.58)
  Day 4 | 67.4 (7.89) | 65.6 (9.37)
  Day 5 | 64.4 (6.97) | 66.9 (8.39)

75. Secondary Outcome: Absolute Values for Vital Sign: Respiratory Rate-Part 1
Description: Respiratory rate was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Breaths per minute
  Baseline; n=18, 18 | 14.0 (2.66) | 14.9 (1.71)
  Day 2; n=17, 17: number analyzed (Participants) | 17 | 17
  Day 2; n=17, 17 | 13.1 (2.56) | 13.9 (2.69)
  Day 3; n=17, 18: number analyzed (Participants) | 17 | 18
  Day 3; n=17, 18 | 14.7 (2.11) | 15.2 (2.49)
  Day 4; n=18, 18 | 13.9 (2.87) | 14.7 (3.07)
  Day 5; n=18, 18 | 14.0 (2.47) | 14.1 (1.75)

76. Secondary Outcome: Absolute Values for Vital Sign: Temperature-Part 1
Description: Temperature was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Degrees Celsius
  Baseline | 36.24 (0.393) | 36.37 (0.361)
  Day 2 | 36.22 (0.426) | 36.39 (0.407)
  Day 3 | 36.33 (0.420) | 36.22 (0.383)
  Day 4 | 36.38 (0.402) | 36.35 (0.385)
  Day 5 | 36.21 (0.555) | 36.27 (0.324)

77. Secondary Outcome: Absolute Values for Vital Signs: DBP and SBP-Part 2
Description: as for outcome 73
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Millimeters of mercury
  SBP, Baseline | 120.8 (17.53) | 115.2 (11.46) | 117.4 (13.01)
  SBP, Day 2 | 117.4 (11.84) | 116.6 (11.32) | 115.7 (11.73)
  SBP, Day 3 | 115.8 (10.63) | 117.2 (11.47) | 116.6 (12.36)
  SBP, Day 4 | 119.0 (12.75) | 115.4 (11.14) | 118.0 (16.87)
  SBP, Day 5 | 118.2 (12.92) | 115.8 (12.76) | 118.0 (13.18)
  DBP, Baseline | 74.8 (10.44) | 71.4 (9.62) | 71.8 (7.51)
  DBP, Day 2 | 72.5 (9.26) | 74.2 (9.83) | 71.1 (7.48)
  DBP, Day 3: number analyzed (Participants) | 7 | 5 | 7
  DBP, Day 3 | 72.9 (7.57) | 72.9 (9.24) | 72.4 (7.53)
  DBP, Day 4 | 71.9 (6.94) | 73.5 (8.32) | 70.5 (9.26)
  DBP, Day 5 | 72.0 (8.61) | 72.3 (7.64) | 68.7 (9.18)

78. Secondary Outcome: Absolute Values for Vital Sign: Pulse Rate-Part 2
Description: as for outcome 74
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Beats per minute
  Baseline | 65.4 (12.47) | 64.1 (7.70) | 63.8 (7.85)
  Day 2 | 66.9 (12.76) | 64.0 (10.66) | 64.1 (7.94)
  Day 3 | 66.7 (11.28) | 64.9 (14.16) | 67.4 (11.04)
  Day 4 | 70.8 (12.90) | 68.2 (11.25) | 72.6 (12.36)
  Day 5 | 67.6 (11.19) | 69.1 (9.11) | 69.6 (13.99)

79. Secondary Outcome: Absolute Values for Vital Sign: Respiratory Rate-Part 2
Description: as for outcome 75
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Breaths per minute
  Baseline | 14.8 (1.20) | 15.3 (2.02) | 13.8 (2.27)
  Day 2 | 14.3 (2.27) | 15.4 (1.64) | 14.2 (2.36)
  Day 3 | 15.0 (2.00) | 14.5 (1.98) | 14.2 (2.18)
  Day 4 | 14.9 (2.38) | 14.0 (3.06) | 14.3 (2.22)
  Day 5 | 13.7 (1.63) | 14.5 (1.61) | 14.6 (1.80)

80. Secondary Outcome: Absolute Values for Vital Sign: Temperature-Part 2
Description: as for outcome 76
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Degrees Celsius
  Baseline | 36.24 (0.421) | 36.50 (0.298) | 36.37 (0.483)
  Day 2 | 36.29 (0.476) | 36.40 (0.406) | 36.27 (0.508)
  Day 3 | 36.33 (0.351) | 36.37 (0.425) | 36.29 (0.419)
  Day 4 | 36.37 (0.404) | 36.37 (0.378) | 36.38 (0.495)
  Day 5 | 36.34 (0.345) | 36.49 (0.375) | 36.51 (0.459)

81. Secondary Outcome: Change From Baseline in Vital Signs: SBP and DBP-Part 1
Description: Blood pressure was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Millimeters of mercury
  SBP; Day 2 | -4.5 (7.52) | -2.3 (7.22)
  SBP; Day 3 | -4.7 (9.63) | -4.1 (9.63)
  SBP; Day 4 | -6.1 (7.45) | -3.4 (10.18)
  SBP; Day 5 | -6.1 (7.49) | -3.6 (11.37)
  DBP; Day 2: number analyzed (Participants) | 9 | 9
  DBP; Day 2 | -2.0 (6.82) | -2.2 (5.78)
  DBP; Day 3 | -1.7 (7.46) | -4.3 (4.80)
  DBP; Day 4 | -1.9 (6.98) | -4.7 (6.99)
  DBP; Day 5 | -2.1 (7.46) | -4.6 (7.17)

82. Secondary Outcome: Change From Baseline in Vital Sign: Pulse Rate-Part 1
Description: as for outcome 74
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Beats per minute
  Day 2 | 1.1 (5.76) | 2.2 (7.50)
  Day 3 | 1.8 (8.20) | 2.4 (7.41)
  Day 4 | 1.7 (6.93) | -0.6 (7.88)
  Day 5 | -1.3 (5.46) | 0.8 (10.70)

83. Secondary Outcome: Change From Baseline in Vital Sign: Respiratory Rate-Part 1
Description: Respiratory rate was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is defined as the latest predose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Breaths per minute
  Day 2; n=17, 17: number analyzed (Participants) | 17 | 17
  Day 2; n=17, 17 | -1.1 (3.47) | -0.8 (3.00)
  Day 3; n=17, 18: number analyzed (Participants) | 17 | 18
  Day 3; n=17, 18 | 0.6 (2.62) | 0.3 (3.58)
  Day 4; n=18, 18 | -0.1 (2.78) | -0.2 (3.35)
  Day 5; n=18, 18 | 0.0 (2.74) | -0.8 (2.76)

84. Secondary Outcome: Change From Baseline in Vital Sign: Temperature-Part 1
Description: Temperature was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is defined as the latest predose assessment with a non-missing value, including those from unscheduled visits, within each treatment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Degrees Celsius
  Day 2 | -0.03 (0.329) | 0.02 (0.472)
  Day 3 | 0.09 (0.442) | -0.15 (0.444)
  Day 4 | 0.13 (0.452) | -0.02 (0.458)
  Day 5 | -0.04 (0.501) | -0.11 (0.330)

85. Secondary Outcome: Change From Baseline in Vital Signs: SBP and DBP-Part 2
Description: as for outcome 81
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Millimeters of mercury
  SBP, Day 2 | -3.5 (10.50) | 1.5 (6.59) | -1.7 (7.65)
  SBP, Day 3 | -5.1 (12.99) | 2.1 (7.74) | -0.9 (9.11)
  SBP, Day 4 | -1.9 (12.28) | 0.3 (6.10) | 0.6 (9.95)
  SBP, Day 5 | -2.6 (11.23) | 0.7 (8.28) | 0.6 (7.71)
  DBP, Day 2 | -2.4 (6.10) | 2.8 (5.07) | -0.7 (4.90)
  DBP, Day 3: number analyzed (Participants) | 7 | 5 | 7
  DBP, Day 3 | -1.9 (6.40) | 1.5 (7.83) | 0.6 (4.95)
  DBP, Day 4 | -2.9 (8.53) | 2.2 (6.27) | -1.3 (6.63)
  DBP, Day 5 | -2.9 (6.19) | 0.9 (6.99) | -3.0 (7.92)

86. Secondary Outcome: Change From Baseline in Vital Sign: Pulse Rate-Part 2
Description: Pulse rate was assessed in the semi-recumbent position with a completely automated device, preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is defined as the average of the triplicate predose assessments within each treatment. Change from Baseline was calculated as post-dose visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Beats per minute
  Day 2 | 1.5 (7.39) | -0.1 (8.02) | 0.3 (4.72)
  Day 3 | 1.3 (9.69) | 0.9 (13.16) | 3.7 (6.59)
  Day 4 | 5.4 (10.17) | 4.1 (9.64) | 8.9 (8.21)
  Day 5 | 2.2 (6.39) | 5.0 (8.37) | 5.9 (8.43)

87. Secondary Outcome: Change From Baseline in Vital Sign: Respiratory Rate-Part 2
Description: as for outcome 83
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Breaths per minute
  Day 2 | -0.5 (2.24) | 0.1 (2.62) | 0.4 (2.58)
  Day 3 | 0.2 (2.42) | -0.7 (2.42) | 0.4 (3.61)
  Day 4 | 0.1 (2.20) | -1.3 (3.72) | 0.5 (2.27)
  Day 5 | -1.1 (1.77) | -0.7 (1.91) | 0.8 (2.86)

88. Secondary Outcome: Change From Baseline in Vital Sign: Temperature-Part 2
Description: as for outcome 84
Time Frame: Baseline (Day 1, pre-dose), Days 2, 3, 4 and 5
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 19 | 21
Degrees Celsius
  Day 2 | 0.05 (0.477) | -0.10 (0.325) | -0.10 (0.390)
  Day 3 | 0.09 (0.302) | -0.13 (0.245) | -0.08 (0.453)
  Day 4 | 0.13 (0.490) | -0.13 (0.268) | 0.01 (0.399)
  Day 5 | 0.10 (0.426) | -0.01 (0.375) | 0.15 (0.437)

89. Secondary Outcome: Lag Time for Absorption (Tlag) for GSK3640254-Part 1
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Hours | 0.528 (0.7568) | 0.139 (0.4132)

90. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) for GSK3640254-Part 1
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Hours | 26.247 (17.6) | 26.185 (17.2)

91. Secondary Outcome: Apparent Oral Clearance (CL/F) for GSK3640254-Part 1
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Liters per hour | 5.413 (42.7) | 5.423 (40.3)

92. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for GSK3640254-Part 1
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Liters | 205.0 (40.0) | 204.9 (43.0)

93. Secondary Outcome: Plasma Concentration of GSK3640254-Part 1
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Concentration Population comprised of all participants who underwent plasma PK sampling and had evaluable PK assay results.
Measure: Median (Full Range); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets
Number analyzed (Participants) | 18 | 18
Nanograms per milliliter
  pre-dose | 1.910 [0 to 44.1] | 1.580 [0 to 31.5]
  1 hour | 6.795 [0 to 80.8] | 81.90 [0 to 842]
  1.5 hours | 26.40 [0 to 421] | 291.0 [0 to 1650]
  2 hours | 104.5 [0 to 991] | 502.5 [28.1 to 2160]
  2.5 hours | 342.5 [0 to 1500] | 804.0 [103 to 2610]
  3 hours | 563.5 [16.7 to 1780] | 965.0 [321 to 2210]
  3.5 hours | 724.0 [44.3 to 1560] | 1105 [482 to 2190]
  4 hours | 798.5 [80.1 to 1660] | 1190 [569 to 1940]
  4.5 hours | 964.5 [135 to 1900] | 1270 [567 to 1890]
  5 hours | 1047 [170 to 1840] | 1195 [479 to 1810]
  6 hours | 1013 [385 to 1750] | 992.0 [437 to 1710]
  8 hours | 981.0 [298 to 1610] | 895.0 [385 to 1500]
  12 hours | 817.0 [253 to 1470] | 787.0 [290 to 1210]
  24 hours | 565.5 [162 to 889] | 582.0 [202 to 887]
  48 hours | 286.0 [81.9 to 483] | 286.0 [121 to 509]
  72 hours | 159.0 [47.3 to 284] | 150.0 [75.1 to 271]
  96 hours | 78.10 [26.0 to 197] | 72.80 [34.0 to 172]

94. Secondary Outcome: Tlag for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 13 | 21
Hours | 0.050 (0.2236) | 0.000 (0.0000) | 0.048 (0.2182)

95. Secondary Outcome: T1/2 for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 10 | 21
Hours | 24.921 (18.0) | 25.669 (12.7) | 24.833 (15.7)

96. Secondary Outcome: CL/F for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 10 | 21
Liter per hour | 4.878 (42.2) | 14.85 (58.2) | 5.417 (35.9)

97. Secondary Outcome: Vz/F for GSK3640254-Part 2
Description: as for outcome 2
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Parameter Population. Only those participants with data available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 10 | 21
Liters | 175.4 (43.4) | 550.1 (66.3) | 194.1 (35.9)

98. Secondary Outcome: Plasma Concentration of GSK3640254-Part 2
Description: Blood samples were collected at indicated time points for PK analysis.
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 12, 24, 48, 72 and 96 hours post-dose
Population: PK Concentration Population. Only those participants with data available at the specified time points were analyzed.
Measure: Median (Full Range); unit: Nanograms per milliliter
Groups:
- Part 2: GSK3640254 200 mg Tablet (Fasted): Participants were administered a single dose of GSK3640254 200 mg tablets, orally under fasted conditions on Day 1 in Period 1 or 2.
Arm/Group | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
Number analyzed (Participants) | 20 | 13 | 21
Nanograms per milliliter
  pre-dose | 6.370 [0 to 31.6] | 0 [0 to 12.8] | NA [NA to 14.7] — Median and lower limit could not be calculated as the values were below the lower limit of quantification.
  1 hour | 39.25 [0 to 504] | 38.70 [7.27 to 268] | 92.30 [0 to 1960]
  1.5 hours | 306.0 [9.18 to 1360] | 84.10 [18.3 to 496] | 239.0 [9.88 to 2000]
  2 hours | 733.0 [37.7 to 1920] | 121.0 [23.9 to 648] | 574.0 [27.0 to 1790]
  2.5 hours | 1075 [193 to 2320] | 194.0 [31.0 to 831] | 684.0 [65.0 to 1770]
  3 hours | 1195 [434 to 2320] | 270.0 [34.1 to 1050] | 724.0 [125 to 2040]
  3.5 hours | 1250 [525 to 2310] | 326.0 [40.0 to 1260] | 785.0 [212 to 2070]
  4 hours | 1305 [607 to 2590] | 358.0 [58.9 to 1270] | 833.0 [230 to 1910]
  4.5 hours | 1245 [636 to 2330] | 324.0 [77.4 to 1480] | 866.0 [272 to 1630]
  5 hours | 1275 [590 to 2470] | 322.0 [71.7 to 1420] | 845.0 [355 to 1620]
  6 hours | 1195 [528 to 2450] | 290.0 [75.8 to 1350] | 968.0 [562 to 1440]
  8 hours | 950.5 [457 to 2110] | 255.0 [57.9 to 1160] | 845.0 [427 to 1370]
  12 hours | 773.0 [363 to 1730] | 217.0 [50.6 to 903] | 734.0 [376 to 1420]
  24 hours | 627.5 [256 to 1150] | 177.0 [49.9 to 722] | 580.0 [276 to 1070]
  48 hours | 335.5 [123 to 533] | 98.60 [35.4 to 327] | 287.0 [149 to 683]
  72 hours | 171.5 [57.7 to 292] | 52.50 [28.3 to 153] | 145.0 [68.0 to 375]
  96 hours | 79.75 [26.4 to 203] | 31.30 [14.8 to 80.7] | 62.20 [35.9 to 224]

ADVERSE EVENTS:
Time Frame: Up to Day 12 for Part 1 and up to Day 19 for Part 2
Description: AEs and SAEs were collected in the Safety Population which comprised of all participants who received at least 1 dose of study medication. Data is presented treatment-wise.
Arm/Group | Part 1: GSK3640254 200 mg Capsules | Part 1: GSK3640254 200 mg Tablets | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) | Part 2: GSK3640254 200 mg Tablet (Fasted) | Part 2: GSK3640254 200 mg Tablet (High Fat)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/20 | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/20 | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/18 | 1/18 | 0/20 | 0/19 | 2/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK3640254 200 mg Capsules (N=18) | Part 1: GSK3640254 200 mg Tablets (N=18) | Part 2: GSK3640254 200 mg Tablet (Moderate Fat) (N=20) | Part 2: GSK3640254 200 mg Tablet (Fasted) (N=19) | Part 2: GSK3640254 200 mg Tablet (High Fat) (N=21)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04263142/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT04263142/SAP_001.pdf